CLINICAL TRIAL: NCT03622593
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab (RO6867461) in Patients With Diabetic Macular Edema (RHINE)
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab (RO6867461) in Participants With Diabetic Macular Edema
Acronym: RHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR40398; 2017-005105-12 (EudraCT Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept; faricimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: Faricimab 6 mg Q8W (Experimental): Participants randomized to Arm A received 6 milligrams (mg) faricimab intravitreal (IVT) injections once every 4 weeks (Q4W) to Week 20, followed by 6 mg faricimab IVT injections once every 8 weeks (Q8W) to Week 96, followed by the final study visit at Week 100.
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- B: Faricimab 6 mg PTI (Experimental): Participants randomized to Arm B received 6 milligrams (mg) faricimab intravitreal (IVT) injections Q4W to at least Week 12, followed by a personalized treatment interval (PTI) dosing of 6 mg faricimab IVT injections up to once every 16 weeks (Q16W) through Week 96, followed by the final study visit at Week 100.
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- C: Aflibercept 2 mg Q8W (Active Comparator): Participants randomized to Arm C received 2 milligrams (mg) aflibercept intravitreal (IVT) injections Q4W to Week 16, followed by 2 mg aflibercept IVT injections Q8W to Week 96, followed by the final study visit at Week 100.
  Interventions: Drug: Aflibercept; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Aflibercept — Aflibercept 2 mg was administered by intravitreal (IVT) injection into the study eye once every 8 weeks (Q8W).
  Other Names: Eylea
  Arms: C: Aflibercept 2 mg Q8W
Drug: Faricimab — Faricimab 6 mg was administered by IVT injection into the study eye either once every 8 weeks (Q8W) in arm A or according to a personalized treatment interval (PTI) in arm B.
  Other Names: VABYSMO™; RO6867461; RG7716
  Arms: A: Faricimab 6 mg Q8W; B: Faricimab 6 mg PTI
Procedure: Sham Procedure — The sham is a procedure that mimics an IVT injection and involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It was administered to participants in all three treatments arms at applicable visits to maintain masking among treatment arms.

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of faricimab administered at 8-week intervals or as specified in the protocol following treatment initiation, compared with aflibercept once every 8 weeks (Q8W), in participants with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of diabetes mellitus (Type 1 or Type 2)
* Hemoglobin A1c (HbA1c) of less than or equal to (≤)10% within 2 months prior to Day 1
* Macular thickening secondary to diabetic macular edema (DME) involving the center of the fovea
* Decreased visual acuity attributable primarily to DME
* Ability and willingness to undertake all scheduled visits and assessments
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 3 months after the final dose of study treatment

Exclusion Criteria:

* Currently untreated diabetes mellitus or previously untreated patients who initiated oral or injectable anti-diabetic medication within 3 months prior to Day 1
* Uncontrolled blood pressure, defined as a systolic value greater than (>)180 millimeters of mercury (mmHg) and/or a diastolic value >100 mmHg while a patient is at rest
* Currently pregnant or breastfeeding, or intend to become pregnant during the study
* Treatment with panretinal photocoagulation or macular laser within 3 months prior to Day 1 to the study eye
* Any intraocular or periocular corticosteroid treatment within 6 months prior to Day 1 to the study eye
* Prior administration of IVT faricimab in either eye
* Active intraocular or periocular infection or active intraocular inflammation in the study eye
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision in the study eye
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than DME in the study eye
* Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (188):
- United States (50):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Northwest Arkansas Retina Associates, Springdale, Arkansas
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retinal Consultants Med Group, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California
  - Bay Area Retina Associates, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Prairie Retina Center, Springfield, Illinois
  - Retina Specialists, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - New York University, New York, New York
  - Ophthalmic Cons of Long Island, Oceanside, New York
  - Retina Assoc of Western NY, Rochester, New York
  - University of Rochester Flaum Eye Institute, Rochester, New York
  - The Retina Consultants, Slingerlands, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Retina Consultants Of Carolina, Greenville, South Carolina
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Center of Texas, Southlake, Texas
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Pacific Northwest Retina, Silverdale, Washington
- Argentina (6):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Fundacion Zambrano, CABA
  - Oftalmos, Capital Federal
  - Oftar, Mendoza
  - Centro Oftalmólogos Especialistas, Rosario
  - Grupo Laser Vision, Rosario
- Australia (7):
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Brazil (9):
  - Hospital de Olhos de Aparecida - HOA, Aparecida de Goiânia, Goiás
  - Centro Brasileiro de Cirurgia, Goiânia, Goiás
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP*X, São Paulo, São Paulo
  - CEMAPE - Centro Médico, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
  - Hosp de Olhos de Sorocaba, Sorocaba, São Paulo
- Canada (10):
  - Calgary Retina Consultants, Calgary, Alberta
  - University of British Columbia - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - QEII - HSC Department of Ophthalmology, Halifax, Nova Scotia
  - Ivey Eye Institute, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - University Health Network Toronto Western Hospital, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
- China (15):
  - Beijing Friendship Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Southwest Hospital , Third Military Medical University, Chongqing
  - Army Medical Center of PLA(Daping Hospital), Chongqing
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The Affiliated Eye Hospital of Nanjing Medical University, Nanjing
  - Shanghai Tenth People's Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Wuxi No.2 People's Hospital, Wuxi
- Czechia (5):
  - FN Hradec Králové, O?ní klinika, Hradec Králové
  - Faculty Hospital Ostrava, Ostrava
  - Faculty Hospital Kralovske Vinohrady, Prague
  - AXON Clinical, Prague
  - Nemocnice Sokolov, Sokolov
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Sjællands Universitetshospital, Roskilde, Roskilde
- France (3):
  - Chi De Creteil, Créteil
  - Centre Ophtalmologique, Paris
  - Centres Ophtalmologique St Exupéry, Saint-Cyr-sur-Loire
- Germany (7):
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Augenheilkunde, Dresden
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Magdeburg A.ö.R., Universitätsaugenklinik, Magdeburg
  - LMU Klinikum der Universität, Augenklinik, München
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Würzburg, Augenklinik und Poliklinik, Würzburg
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - Hong Kong Eye Hospital, Mong Kok
- Hungary (4):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Szemeszet KR, Budapest
  - Semmelweis Egyetem Szemészeti Vizsgálóhely, Budapest
  - Bajcsy-Zsilinszky Hospital, Budapest
- Italy (5):
  - Fondazione Ptv Policlinico Tor Vergata Di Roma, Rome, Lazio
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Nuovo Ospedale S. Chiara - A.O.U.P Presidio Ospedaliero di Cisanello, Pisa, Tuscany
  - Ospedale Classificato Equiparato Sacro Cuore Don Calabria, Negrar, Veneto
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Veneto
- Poland (8):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Specjalistyczny O?rodek Okulistyczny Oculomedica, Bydgoszcz
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Niepubliczny Zaklad Opieki Zdrowotnej PRYZMAT-OKULISTYKA, Gliwice
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzia? Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Osrodek Chirurgii Oka prof. Zagorskiego Rzeszow, Rzeszów
  - Caminomed, Tarnowskie Góry
  - Centrum Zdrowia MDM, Warsaw
- Portugal (4):
  - Hospital de Braga, Braga
  - AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra
  - Espaco Medico Coimbra, Coimbra
  - Hospital de Santa Maria, Lisbon
- Russia (4):
  - Intersec Research and Technology Complex ?Eye Microsurgery? n.a. S.N. Fyodorov, Cheboksary, Mariy-El Republic
  - Clinics of Eye Diseases, LLC, Kazan', Tatarstan Republic
  - ?Intersec. Research and Technology Complex ?Eye Microsurgery? n a Fyodorov Irkutsk branch, Irkutsk
  - ?Intersec Research and Technology Complex Eye Microsurgery n a Fyodorov Novosibirsk Branch, Novosibirsk
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center., Seoul
- Spain (9):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Oftalvist Valencia, Burjassot, Valencia
  - Hospital dos de maig, Barcelona
  - Clinica Baviera, Madrid
  - Fisabio-Ofalmologia Medica, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
- Vista Klinik Ophthalmologische Klinik, Binningen, Switzerland
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Maharaj Nakorn ChiangMai Hospital, Chiang Mai
- Turkey (Türkiye) (4):
  - Ankara University Medical Faculty; Department of Ophthalmology, Ankara
  - Ankara Baskent University Medical Faculty; Department of Ophthalmology, Ankara
  - Beyoglu Goz Training and Research Hospital; Department Of Ophthalmology, Istanbul
  - Kocaeli Üniversitesi T?p Fakültesi; Department of Ophthalmology, Kocaeli
- United Kingdom (18):
  - Barnet Hospital, Barnet
  - Bradford Royal Infirmary, Bradford
  - University Hospitals Bristol NHS Foundation Trust, Bristol Eye Hospital, Bristol
  - Belfast Health and Social Care Trust, ROYAL VICTORIA HOSPITAL, Bristol
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Frimley Park Hospital, Frimley
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Royal Free Hospital, London
  - Kings College Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Sunderland Eye Infirmary, Sunderland
  - Hillingdon Hospital, Uxbridge

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Result] Wong TY, Haskova Z, Asik K, Baumal CR, Csaky KG, Eter N, Ives JA, Jaffe GJ, Korobelnik JF, Lin H, Murata T, Ruamviboonsuk P, Schlottmann PG, Seres AI, Silverman D, Sun X, Tang Y, Wells JA, Yoon YH, Wykoff CC; YOSEMITE and RHINE Investigators. Faricimab Treat-and-Extend for Diabetic Macular Edema: Two-Year Results from the Randomized Phase 3 YOSEMITE and RHINE Trials. Ophthalmology. 2024 Jun;131(6):708-723. doi: 10.1016/j.ophtha.2023.12.026. Epub 2023 Dec 28. PMID 38158159
- [Derived] Sheth VS, Schlottmann P, Lai TYY, Abreu F, Chang A, Eter N, Gibson K, Hu AY, Korobelnik JF, Kotak A, Kotecha A, O'Leary OE, Pearce I, Sim DA, Sun JK, Tang Y, Khanani AM. Four-Year Outcomes of Faricimab in Diabetic Macular Edema: Results From the RHONE-X Extension Trial. Ophthalmology. 2026 Jan 12:S0161-6420(26)00004-7. doi: 10.1016/j.ophtha.2026.01.001. Online ahead of print. PMID 41534798
- [Derived] Jaffe GJ, Deak G, Gibson K, Khurana RN, Nudleman E, Ogura Y, Schmidt-Erfurth U, Wang T, Westenskow PD, Wong D, Yiu G, Willis JR. IMPACT OF FARICIMAB VERSUS AFLIBERCEPT ON EPIRETINAL MEMBRANE FORMATION OVER 2 YEARS IN PATIENTS WITH DIABETIC MACULAR EDEMA IN THE PHASE 3 YOSEMITE AND RHINE TRIALS. Retina. 2025 Nov 1;45(11):2003-2011. doi: 10.1097/IAE.0000000000004572. PMID 40668667
- [Derived] Chakravarthy U, Chaudhary V, Sadda SR, Tan CS, Vujosevic S, Fauser S, Gibson K, Glittenberg C, Holekamp N, Lanza B, Maunz A, Willis JR, Singh RP. Effect of Faricimab versus Aflibercept on Hyperreflective Foci in Patients with Diabetic Macular Edema from the YOSEMITE/RHINE Trials. Ophthalmol Sci. 2025 Apr 19;5(5):100798. doi: 10.1016/j.xops.2025.100798. eCollection 2025 Sep-Oct. PMID 40496217
- [Derived] Goldberg RA, Mar FA, Csaky K, Amador M, Khanani AM, Gibson K, Kolomeyer AM, Sim DA, Murata T, Wang T, Udaondo P, Souverain A, Shildkrot YE, Vujosevic S, Nudleman E, Sivaprasad S. Resolution of Angiographic Macular Leakage with Faricimab versus Aflibercept in Patients with Diabetic Macular Edema in YOSEMITE/RHINE. Ophthalmol Retina. 2025 Jun;9(6):515-526. doi: 10.1016/j.oret.2024.11.015. Epub 2024 Nov 22. PMID 39580145
- [Derived] Stockwell AD, Chang MC, Mahajan A, Forrest W, Anegondi N, Pendergrass RK, Selvaraj S, Reeder J, Wei E, Iglesias VA, Creps NM, Macri L, Neeranjan AN, van der Brug MP, Scales SJ, McCarthy MI, Yaspan BL. Multi-ancestry GWAS analysis identifies two novel loci associated with diabetic eye disease and highlights APOL1 as a high risk locus in patients with diabetic macular edema. PLoS Genet. 2023 Aug 16;19(8):e1010609. doi: 10.1371/journal.pgen.1010609. eCollection 2023 Aug. PMID 37585454
- [Derived] Shimura M, Kitano S, Ogata N, Mitamura Y, Oh H, Ochi H, Ohsawa S, Hirakata A; YOSEMITE and RHINE Investigators. Efficacy, durability, and safety of faricimab with extended dosing up to every 16 weeks in Japanese patients with diabetic macular edema: 1-year results from the Japan subgroup of the phase 3 YOSEMITE trial. Jpn J Ophthalmol. 2023 May;67(3):264-279. doi: 10.1007/s10384-023-00979-8. Epub 2023 Mar 10. PMID 36897413
- [Derived] Eter N, Singh RP, Abreu F, Asik K, Basu K, Baumal C, Chang A, Csaky KG, Haskova Z, Lin H, Ruiz CQ, Ruamviboonsuk P, Silverman D, Wykoff CC, Willis JR. YOSEMITE and RHINE: Phase 3 Randomized Clinical Trials of Faricimab for Diabetic Macular Edema: Study Design and Rationale. Ophthalmol Sci. 2021 Dec 30;2(1):100111. doi: 10.1016/j.xops.2021.100111. eCollection 2022 Mar. PMID 36246184
- [Derived] Wykoff CC, Abreu F, Adamis AP, Basu K, Eichenbaum DA, Haskova Z, Lin H, Loewenstein A, Mohan S, Pearce IA, Sakamoto T, Schlottmann PG, Silverman D, Sun JK, Wells JA, Willis JR, Tadayoni R; YOSEMITE and RHINE Investigators. Efficacy, durability, and safety of intravitreal faricimab with extended dosing up to every 16 weeks in patients with diabetic macular oedema (YOSEMITE and RHINE): two randomised, double-masked, phase 3 trials. Lancet. 2022 Feb 19;399(10326):741-755. doi: 10.1016/S0140-6736(22)00018-6. Epub 2022 Jan 24. PMID 35085503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Started (Intent-to-Treat (ITT) Population) | 317 | 319 | 315
Received at Least One Dose of Study Drug (Safety-Evaluable Population) | 317 | 319 | 314
Completed up to Week 56 (Primary Completion Date Cutoff) | 298 | 312 | 299
Completed | 275 | 288 | 267
Not Completed | 42 | 31 | 48
Not completed — Withdrawal by Subject | 11 | 9 | 13
Not completed — Death | 12 | 9 | 10
Not completed — Lost to Follow-up | 11 | 5 | 8
Not completed — Adverse Event | 4 | 5 | 6
Not completed — Physician Decision | 2 | 1 | 6
Not completed — Other | 2 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants (951) comprises the Intent-to-Treat (ITT) Population, which includes all global participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W | Total
Number analyzed (Participants) | 317 | 319 | 315 | 951
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Years
    ITT Population | 62.5 (10.1) | 61.6 (10.1) | 62.3 (10.1) | 62.2 (10.1)
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population | 62.5 (9.9) | 61.3 (10.3) | 62.5 (10.0) | 62.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: Female | 123 | 120 | 129 | 372
    ITT Population: Male | 194 | 199 | 186 | 579
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: Female | 100 | 94 | 97 | 291
    Treatment-Naive Population: Male | 154 | 161 | 151 | 466
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: Hispanic or Latino | 56 | 78 | 67 | 201
    ITT Population: Not Hispanic or Latino | 252 | 232 | 240 | 724
    ITT Population: Unknown or Not Reported | 9 | 9 | 8 | 26
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: Hispanic or Latino | 42 | 57 | 54 | 153
    Treatment-Naive Population: Not Hispanic or Latino | 204 | 190 | 188 | 582
    Treatment-Naive Population: Unknown or Not Reported | 8 | 8 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: American Indian or Alaska Native | 0 | 0 | 1 | 1
    ITT Population: Asian | 34 | 36 | 32 | 102
    ITT Population: Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
    ITT Population: Black or African American | 18 | 23 | 24 | 65
    ITT Population: White | 250 | 249 | 253 | 752
    ITT Population: More than one race | 2 | 1 | 0 | 3
    ITT Population: Unknown or Not Reported | 11 | 10 | 5 | 26
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Treatment-Naive Population: Asian | 26 | 29 | 25 | 80
    Treatment-Naive Population: Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
    Treatment-Naive Population: Black or African American | 16 | 20 | 17 | 53
    Treatment-Naive Population: White | 197 | 197 | 201 | 595
    Treatment-Naive Population: More than one race | 2 | 1 | 0 | 3
    Treatment-Naive Population: Unknown or Not Reported | 11 | 8 | 5 | 24
Number of Participants by Previous Treatment Status with Intravitreal Anti-VEGF Agents [Count of Participants; unit: Participants] — The Treatment-Naive Population was defined as all participants randomized in the study who had not received any intravitreal (IVT) anti-VEGF agents in the study eye prior to randomization.
  Participants
    Treatment-Naive | 254 | 255 | 248 | 757
    Previously Treated | 63 | 64 | 67 | 194
Region of Enrollment [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: United States and Canada | 110 | 111 | 109 | 330
    ITT Population: Asia | 29 | 29 | 26 | 84
    ITT Population: Rest of the World | 178 | 179 | 180 | 537
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: United States and Canada | 87 | 88 | 84 | 259
    Treatment-Naive Population: Asia | 23 | 24 | 21 | 68
    Treatment-Naive Population: Rest of the World | 144 | 143 | 143 | 430
Number of Participants by the Eye Chosen as the Study Eye (Left or Right) [Count of Participants; unit: Participants] — Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: Left Eye | 156 | 168 | 146 | 470
    ITT Population: Right Eye | 161 | 151 | 169 | 481
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: Left Eye | 128 | 136 | 117 | 381
    Treatment-Naive Population: Right Eye | 126 | 119 | 131 | 376
Baseline Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye [Mean (Standard Deviation); unit: ETDRS Letters] — Best corrected visual acuity (BCVA) was measured at a starting test distance of 4 meters using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity. Population: The ITT Population (951) includes all global participants randomized in the study. The Treatment-Naive Population (757), ITT subset, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization. 3 participants (1 in Arm A and 2 in Arm B) were excluded for missing or invalid BCVA values.
  ETDRS Letters
    ITT Population: number analyzed (Participants) | 316 | 317 | 315 | 948
    ITT Population | 61.9 (10.1) | 62.5 (9.3) | 62.1 (9.4) | 62.1 (9.6)
    Treatment-Naive Population: number analyzed (Participants) | 253 | 253 | 248 | 754
    Treatment-Naive Population | 62.1 (10.1) | 62.8 (9.3) | 62.6 (9.2) | 62.5 (9.5)
Number of Participants by the Baseline BCVA Letter Score Categories in the Study Eye [Count of Participants; unit: Participants] — Best corrected visual acuity (BCVA) was measured at a starting test distance of 4 meters using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity. Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: ≤38 Letters | 14 | 11 | 9 | 34
    ITT Population: 39 to 63 Letters | 128 | 132 | 132 | 392
    ITT Population: ≥64 Letters | 174 | 174 | 174 | 522
    ITT Population: Missing/Invalid BCVA | 1 | 2 | 0 | 3
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: ≤38 Letters | 10 | 8 | 5 | 23
    Treatment-Naive Population: 39 to 63 Letters | 100 | 103 | 100 | 303
    Treatment-Naive Population: ≥64 Letters | 143 | 142 | 143 | 428
    Treatment-Naive Population: Missing/Invalid BCVA | 1 | 2 | 0 | 3
Number of Participants by Baseline Diabetic Retinopathy Severity (DRS) Status in the Study Eye [Count of Participants; unit: Participants] — The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by the central reading center. Population: The ITT and Treatment-Naive (TN) Populations are grouped according to treatment assigned at randomization. The ITT Population (951) includes all global participants randomized in the study. The TN Population (757), a subset of ITT, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization.
  Participants
    ITT Population: 1 - Diabetic Retinopathy (DR) Absent | 2 | 4 | 1 | 7
    ITT Population: 2 - DR Questionable / Microaneurysms Only | 3 | 10 | 6 | 19
    ITT Population: 3 - Mild Non-Proliferative Diabetic Retinopathy (NPDR) | 90 | 92 | 94 | 276
    ITT Population: 4 - Moderate NPDR | 88 | 72 | 79 | 239
    ITT Population: 5 - Moderately Severe NPDR | 59 | 63 | 54 | 176
    ITT Population: 6 - Severe NPDR | 50 | 36 | 51 | 137
    ITT Population: 7 - Mild Proliferative Diabetic Retinopathy (PDR) | 12 | 26 | 11 | 49
    ITT Population: 8 - Moderate PDR | 6 | 10 | 6 | 22
    ITT Population: 9 - High Risk PDR (DRS Level 71) | 2 | 1 | 3 | 6
    ITT Population: 10 - High Risk PDR (DRS Level 75) | 0 | 0 | 0 | 0
    ITT Population: 11 - Advanced PDR (DRS Level 81) | 0 | 0 | 0 | 0
    ITT Population: 12 - Advanced PDR (DRS Level 85) | 0 | 0 | 0 | 0
    ITT Population: Cannot Grade | 2 | 5 | 5 | 12
    ITT Population: Missing | 3 | 0 | 5 | 8
    Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248 | 757
    Treatment-Naive Population: 1 - Diabetic Retinopathy (DR) Absent | 2 | 3 | 1 | 6
    Treatment-Naive Population: 2 - DR Questionable / Microaneurysms Only | 1 | 8 | 6 | 15
    Treatment-Naive Population: 3 - Mild Non-Proliferative Diabetic Retinopathy (NPDR) | 63 | 66 | 71 | 200
    Treatment-Naive Population: 4 - Moderate NPDR | 74 | 59 | 56 | 189
    Treatment-Naive Population: 5 - Moderately Severe NPDR | 48 | 56 | 43 | 147
    Treatment-Naive Population: 6 - Severe NPDR | 44 | 32 | 47 | 123
    Treatment-Naive Population: 7 - Mild Proliferative Diabetic Retinopathy (PDR) | 11 | 17 | 7 | 35
    Treatment-Naive Population: 8 - Moderate PDR | 5 | 9 | 5 | 19
    Treatment-Naive Population: 9 - High Risk PDR (DRS Level 71) | 2 | 1 | 3 | 6
    Treatment-Naive Population: 10 - High Risk PDR (DRS Level 75) | 0 | 0 | 0 | 0
    Treatment-Naive Population: 11 - Advanced PDR (DRS Level 81) | 0 | 0 | 0 | 0
    Treatment-Naive Population: 12 - Advanced PDR (DRS Level 85) | 0 | 0 | 0 | 0
    Treatment-Naive Population: Cannot Grade | 1 | 4 | 4 | 9
    Treatment-Naive Population: Missing | 3 | 0 | 5 | 8
Baseline Central Subfield Thickness in the Study Eye [Mean (Standard Deviation); unit: microns] — Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by the central reading center. Population: The ITT Population (951) includes all global participants randomized in the study. The Treatment-Naive Population (757), ITT subset, includes randomized participants who had not received any IVT anti-VEGF agents in the study eye before randomization. Nine participants in the ITT (3 per arm) were excluded for missing or ungradable assessments.
  microns
    ITT Population: number analyzed (Participants) | 314 | 316 | 312 | 942
    ITT Population | 466.2 (119.4) | 471.3 (127.0) | 477.3 (129.4) | 471.6 (125.3)
    Treatment-Naive Population: number analyzed (Participants) | 251 | 252 | 248 | 751
    Treatment-Naive Population | 464.6 (117.9) | 473.0 (130.5) | 474.3 (129.5) | 470.6 (126.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded. 97.5% CI is a rounding of 97.52% CI.
Time Frame: From Baseline through Week 56
Population: ITT Population and Treatment-Naive Population
Measure: Mean (97.5% Confidence Interval); unit: ETDRS Letters
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
ETDRS Letters
  ITT Population | 11.8 [10.6 to 13.0] | 10.8 [9.6 to 11.9] | 10.3 [9.1 to 11.4]
  Treatment-Naive Population: number analyzed (Participants) | 254 | 255 | 248
  Treatment-Naive Population | 11.7 [10.4 to 13.0] | 11.2 [9.9 to 12.4] | 10.5 [9.2 to 11.9]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the non-inferiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in adjusted means for the faricimab 6 mg Q8W and the active comparator (aflibercept 2 mg Q8W) arms was greater than -4 letters, then faricimab 6 mg Q8W was considered non-inferior to aflibercept 2 mg Q8W. Non-inferiority was tested one-sided at a significance level of α = 0.0248; Adjusted mean difference = 1.5, 97.5% CI 2-sided [-0.1 to 3.2], Standard Error of Mean 0.73 — The difference in adjusted means was calculated as Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the ITT Population
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the non-inferiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in adjusted means for the faricimab 6 mg PTI and the active comparator (aflibercept 2 mg Q8W) arms was greater than -4 letters, then faricimab 6 mg PTI was considered non-inferior to aflibercept 2 mg Q8W. Non-inferiority was tested one-sided at a significance level of α = 0.0248; Adjusted mean difference = 0.5, 97.5% CI 2-sided [-1.1 to 2.1], Standard Error of Mean 0.73 — The difference in adjusted means was calculated as Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the ITT Population
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.1718, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = 1.1, 97.5% CI 2-sided [-0.7 to 3.0], Standard Error of Mean 0.83 — The difference in adjusted means was calculated as Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.4602, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = 0.6, 97.5% CI 2-sided [-1.2 to 2.4], Standard Error of Mean 0.82 — The difference in adjusted means was calculated as Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.0361, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = 1.5, 97.5% CI 2-sided [-0.1 to 3.2], Standard Error of Mean 0.73 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; Three hypotheses were tested in order for each faricimab arm (Q8W or PTI) separately against the aflibercept arm using a graph-based testing procedure. The analysis presented here is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.4930, Mixed Model for Repeated Measures — Tested at an overall significance level of α = 0.0248; Adjusted mean difference = 0.5, 97.5% CI 2-sided [-1.1 to 2.1], Standard Error of Mean 0.73 — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With a ≥2-Step Diabetic Retinopathy Severity (DRS) Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale (DRSS) at Week 52, ITT and Treatment-Naive Populations
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 97.5% confidence interval (CI) is a rounding of 97.52% CI.
Time Frame: Baseline and Week 52
Population: ITT Population and Treatment-Naive Population. Only participants with non-missing, valid assessments at Baseline and Week 52 were included in the analysis.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 231 | 251 | 238
Percentage of participants
  ITT Population | 44.2 [37.1 to 51.4] | 43.7 [36.8 to 50.7] | 46.8 [39.8 to 53.8]
  Treatment-Naive Population: number analyzed (Participants) | 179 | 198 | 184
  Treatment-Naive Population | 46.9 [38.7 to 55.1] | 45.7 [37.8 to 53.7] | 52.3 [44.2 to 60.4]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This analysis is for the non-inferiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in CMH weighted percentages of participants for the faricimab Q8W and the active comparator (aflibercept Q8W) arms was greater than -10%, then faricimab Q8W was considered non-inferior to aflibercept; Difference in CMH Weighted Percentage = -2.6, 97.5% CI 2-sided [-12.6 to 7.4]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This analysis is for the non-inferiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Non-Inferiority — If the lower bound of the two-sided 97.52% confidence interval for the difference in CMH weighted percentages of participants for the faricimab PTI and the active comparator (aflibercept Q8W) arms was greater than -10%, then faricimab PTI was considered non-inferior to aflibercept; Difference in CMH Weighted Percentage = -3.5, 97.5% CI 2-sided [-13.4 to 6.3]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This analysis is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.3009, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = -5.4, 97.5% CI 2-sided [-16.9 to 6.1]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This analysis is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Superiority; p = 0.1735, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = -6.9, 97.5% CI 2-sided [-18.3 to 4.4]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This analysis is for the superiority of Arm A: Faricimab 6 mg Q8W compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.5757, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = -2.6, 97.5% CI 2-sided [-12.6 to 7.4]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This analysis is for the superiority of Arm B: Faricimab 6 mg PTI compared with Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Superiority; p = 0.4293, Cochran-Mantel-Haenszel — Tested at an overall significance level of α = 0.0248; Difference in CMH Weighted Percentage = -3.5, 97.5% CI 2-sided [-13.4 to 6.3]

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
ETDRS Letters
  Week 4 | 6.1 [5.4 to 6.8] | 6.6 [5.8 to 7.3] | 6.4 [5.7 to 7.1]
  Week 8 | 7.8 [7.0 to 8.5] | 8.1 [7.4 to 8.9] | 7.5 [6.8 to 8.3]
  Week 12 | 8.7 [7.8 to 9.5] | 9.1 [8.2 to 9.9] | 8.5 [7.7 to 9.4]
  Week 16 | 9.9 [9.0 to 10.7] | 9.8 [9.0 to 10.7] | 8.8 [7.9 to 9.6]
  Week 20 | 10.1 [9.2 to 10.9] | 9.5 [8.6 to 10.4] | 8.8 [8.0 to 9.7]
  Week 24 | 10.6 [9.7 to 11.5] | 9.9 [9.0 to 10.8] | 9.3 [8.4 to 10.2]
  Week 28 | 10.7 [9.7 to 11.6] | 10.5 [9.6 to 11.4] | 9.6 [8.7 to 10.5]
  Week 32 | 11.3 [10.3 to 12.3] | 10.2 [9.2 to 11.1] | 9.4 [8.5 to 10.4]
  Week 36 | 11.0 [10.1 to 12.0] | 10.6 [9.6 to 11.6] | 10.4 [9.5 to 11.4]
  Week 40 | 11.4 [10.3 to 12.5] | 10.7 [9.6 to 11.7] | 10.3 [9.2 to 11.3]
  Week 44 | 11.7 [10.7 to 12.7] | 10.9 [9.9 to 11.9] | 10.5 [9.5 to 11.5]
  Week 48 | 11.8 [10.7 to 12.9] | 10.6 [9.5 to 11.7] | 10.1 [9.0 to 11.1]
  Week 52 | 11.6 [10.5 to 12.6] | 10.7 [9.6 to 11.7] | 10.4 [9.3 to 11.4]
  Week 56 | 11.6 [10.4 to 12.8] | 10.6 [9.5 to 11.8] | 9.9 [8.7 to 11.1]
  Week 60 | 11.4 [10.2 to 12.6] | 10.1 [8.9 to 11.3] | 10.1 [8.9 to 11.3]
  Week 64 | 11.6 [10.4 to 12.7] | 10.3 [9.2 to 11.5] | 9.4 [8.2 to 10.6]
  Week 68 | 11.2 [10.0 to 12.3] | 10.1 [9.0 to 11.3] | 10.0 [8.8 to 11.1]
  Week 72 | 11.2 [9.9 to 12.4] | 9.9 [8.8 to 11.1] | 9.4 [8.2 to 10.6]
  Week 76 | 10.6 [9.3 to 11.9] | 9.4 [8.1 to 10.7] | 9.5 [8.2 to 10.8]
  Week 80 | 10.6 [9.2 to 12.0] | 9.5 [8.1 to 10.9] | 9.1 [7.7 to 10.5]
  Week 84 | 9.8 [8.4 to 11.2] | 10.3 [9.0 to 11.7] | 9.6 [8.2 to 11.0]
  Week 88 | 9.8 [8.4 to 11.3] | 10.0 [8.6 to 11.4] | 9.2 [7.7 to 10.6]
  Week 92 | 10.8 [9.3 to 12.2] | 10.2 [8.8 to 11.7] | 9.3 [7.9 to 10.8]
  Week 96 | 11.3 [9.8 to 12.8] | 10.5 [9.1 to 12.0] | 9.0 [7.5 to 10.5]
  Week 100 | 10.7 [9.1 to 12.3] | 9.5 [7.9 to 11.0] | 9.8 [8.2 to 11.4]

4. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Over Time, Treatment-Naive Population
Description: Best-Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline BCVA (continuous), baseline BCVA (<64 vs. ≥64 letters), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: Treatment-Naive (TN) Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. One participant in Arm B: Faricimab 6 mg PTI was excluded from the TN Population for the final analysis due to a late report of prior anti-VEGF treatment.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
ETDRS Letters
  Week 4 | 6.0 [5.2 to 6.9] | 6.7 [5.8 to 7.5] | 6.3 [5.4 to 7.1]
  Week 8 | 7.5 [6.6 to 8.4] | 8.2 [7.3 to 9.1] | 7.3 [6.4 to 8.2]
  Week 12 | 8.7 [7.8 to 9.6] | 9.2 [8.3 to 10.1] | 8.5 [7.6 to 9.5]
  Week 16 | 9.7 [8.8 to 10.7] | 10.0 [9.1 to 10.9] | 8.7 [7.8 to 9.6]
  Week 20 | 10.0 [9.1 to 11.0] | 9.8 [8.8 to 10.7] | 9.0 [8.1 to 10.0]
  Week 24 | 10.6 [9.6 to 11.6] | 10.2 [9.2 to 11.2] | 9.4 [8.4 to 10.4]
  Week 28 | 10.8 [9.8 to 11.8] | 10.8 [9.8 to 11.8] | 9.9 [8.9 to 10.9]
  Week 32 | 11.2 [10.1 to 12.3] | 10.3 [9.2 to 11.4] | 9.9 [8.8 to 11.0]
  Week 36 | 10.8 [9.7 to 11.9] | 10.9 [9.8 to 12.0] | 10.5 [9.3 to 11.6]
  Week 40 | 11.3 [10.2 to 12.5] | 11.2 [10.0 to 12.3] | 10.6 [9.5 to 11.8]
  Week 44 | 11.5 [10.4 to 12.7] | 11.2 [10.1 to 12.3] | 11.1 [9.9 to 12.2]
  Week 48 | 11.4 [10.2 to 12.7] | 10.9 [9.7 to 12.1] | 10.5 [9.3 to 11.7]
  Week 52 | 11.7 [10.5 to 12.8] | 11.1 [9.9 to 12.2] | 10.7 [9.5 to 11.9]
  Week 56 | 11.4 [10.0 to 12.8] | 11.0 [9.6 to 12.3] | 10.0 [8.6 to 11.4]
  Week 60 | 11.4 [10.0 to 12.7] | 10.5 [9.2 to 11.8] | 10.1 [8.8 to 11.5]
  Week 64 | 11.6 [10.2 to 12.9] | 10.5 [9.2 to 11.8] | 9.5 [8.2 to 10.8]
  Week 68 | 11.2 [9.9 to 12.5] | 10.3 [9.0 to 11.6] | 10.0 [8.7 to 11.3]
  Week 72 | 11.1 [9.7 to 12.5] | 10.1 [8.8 to 11.5] | 9.6 [8.2 to 10.9]
  Week 76 | 10.6 [9.0 to 12.1] | 9.7 [8.2 to 11.2] | 9.5 [8.0 to 11.1]
  Week 80 | 10.9 [9.4 to 12.5] | 10.0 [8.5 to 11.5] | 9.3 [7.8 to 10.9]
  Week 84 | 9.9 [8.4 to 11.5] | 10.8 [9.3 to 12.3] | 9.6 [8.0 to 11.1]
  Week 88 | 9.6 [7.9 to 11.2] | 10.2 [8.6 to 11.8] | 9.4 [7.8 to 11.1]
  Week 92 | 10.4 [8.8 to 12.1] | 10.6 [9.0 to 12.2] | 9.6 [7.9 to 11.2]
  Week 96 | 10.6 [8.9 to 12.3] | 10.9 [9.2 to 12.5] | 9.0 [7.3 to 10.7]
  Week 100 | 10.4 [8.5 to 12.2] | 10.0 [8.2 to 11.7] | 9.8 [7.9 to 11.6]

5. Secondary Outcome: Percentage of Participants Gaining Greater Than or Equal to (≥)15, ≥10, ≥5, or ≥0 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT Population
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with at least one non-missing, valid assessment at Weeks 48, 52, or 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 268 | 293 | 279
Percentage of participants
  Gaining ≥15 Letters | 33.8 [28.4 to 39.2] | 28.5 [23.6 to 33.3] | 30.3 [25.0 to 35.5]
  Gaining ≥10 Letters | 59.3 [53.6 to 64.9] | 53.0 [47.5 to 58.5] | 53.9 [48.3 to 59.5]
  Gaining ≥5 Letters | 81.8 [77.3 to 86.4] | 77.4 [72.7 to 82.1] | 78.0 [73.3 to 82.7]
  Gaining ≥0 Letters | 92.1 [89.0 to 95.3] | 91.1 [87.8 to 94.3] | 91.4 [88.2 to 94.6]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥15 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 3.5, 95% CI 2-sided [-4.0 to 11.1]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥15 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -2.0, 95% CI 2-sided [-9.1 to 5.2]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥10 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 5.4, 95% CI 2-sided [-2.5 to 13.4]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥10 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -1.1, 95% CI 2-sided [-8.9 to 6.8]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥5 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 3.8, 95% CI 2-sided [-2.7 to 10.3]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥5 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.7, 95% CI 2-sided [-7.3 to 5.9]
Statistical Analysis 7: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥0 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.7, 95% CI 2-sided [-3.8 to 5.2]
Statistical Analysis 8: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants gaining ≥0 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.3, 95% CI 2-sided [-4.9 to 4.2]

6. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. At each timepoint, only participants with non-missing, valid assessments were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 13.4 [9.9 to 17.0] | 10.8 [7.5 to 14.2] | 10.6 [7.3 to 14.0]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 15.2 [11.2 to 19.1] | 16.7 [12.7 to 20.8] | 15.4 [11.5 to 19.4]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 20.7 [16.3 to 25.1] | 22.1 [17.6 to 26.5] | 19.3 [15.0 to 23.6]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 24.4 [19.7 to 29.1] | 24.3 [19.7 to 28.8] | 23.1 [18.5 to 27.7]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 26.7 [21.8 to 31.6] | 21.3 [16.8 to 25.7] | 22.8 [18.3 to 27.4]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 29.8 [24.7 to 34.9] | 24.0 [19.3 to 28.6] | 24.6 [19.8 to 29.3]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 30.1 [25.0 to 35.3] | 26.7 [21.9 to 31.5] | 25.7 [20.7 to 30.6]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 35.9 [30.6 to 41.3] | 27.3 [22.2 to 32.3] | 23.9 [19.1 to 28.7]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 33.8 [28.5 to 39.1] | 32.1 [27.0 to 37.2] | 28.5 [23.5 to 33.5]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 37.8 [32.3 to 43.3] | 30.5 [25.4 to 35.6] | 29.1 [24.0 to 34.2]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 37.1 [31.6 to 42.5] | 30.1 [25.0 to 32.5] | 33.4 [28.0 to 38.7]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 33.0 [27.5 to 38.6] | 29.4 [24.4 to 34.3] | 29.3 [24.1 to 34.4]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 35.0 [29.6 to 40.4] | 31.0 [25.9 to 36.2] | 33.1 [27.7 to 38.5]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 38.8 [33.2 to 44.3] | 29.5 [24.5 to 34.6] | 36.4 [30.7 to 42.0]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 38.0 [32.3 to 43.7] | 30.3 [25.2 to 35.5] | 36.6 [30.9 to 42.3]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 40.3 [34.7 to 45.9] | 29.6 [24.5 to 34.8] | 31.9 [26.5 to 37.3]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 36.9 [31.3 to 42.5] | 31.1 [25.8 to 36.5] | 35.4 [29.8 to 41.0]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 36.8 [31.0 to 42.6] | 30.5 [25.1 to 35.8] | 32.5 [26.9 to 38.0]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 37.1 [31.5 to 42.7] | 31.2 [25.9 to 36.6] | 35.1 [29.4 to 40.8]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 39.6 [33.8 to 45.5] | 30.1 [24.8 to 35.3] | 35.3 [29.6 to 41.1]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 38.5 [32.9 to 44.2] | 30.6 [25.2 to 36.0] | 38.1 [32.4 to 43.9]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 40.4 [34.7 to 46.1] | 29.6 [24.3 to 35.0] | 38.5 [32.6 to 44.3]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 42.3 [36.4 to 48.1] | 34.6 [29.2 to 40.0] | 42.1 [36.0 to 48.2]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 44.2 [38.1 to 50.2] | 34.4 [29.0 to 39.7] | 36.0 [30.1 to 41.8]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 43.1 [37.1 to 49.1] | 31.2 [25.9 to 36.5] | 40.8 [34.8 to 46.9]

7. Secondary Outcome: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 29.1 [24.2 to 34.0] | 26.9 [22.1 to 31.8] | 28.7 [23.8 to 33.6]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 39.7 [34.4 to 45.1] | 41.4 [36.0 to 46.9] | 34.8 [29.6 to 40.0]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 44.8 [39.3 to 50.2] | 46.9 [41.4 to 52.4] | 43.2 [37.7 to 48.8]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 52.5 [46.9 to 58.0] | 51.3 [45.9 to 56.7] | 41.8 [36.3 to 47.3]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 54.0 [48.6 to 59.5] | 50.0 [44.5 to 55.6] | 45.5 [40.0 to 51.0]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 57.0 [51.5 to 62.5] | 52.8 [47.4 to 58.3] | 48.4 [42.9 to 53.9]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 58.3 [52.7 to 63.9] | 51.3 [45.8 to 56.8] | 51.7 [46.1 to 57.3]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 60.1 [54.4 to 65.8] | 50.9 [45.2 to 56.6] | 52.5 [46.8 to 58.1]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 58.6 [52.9 to 64.2] | 57.3 [51.7 to 62.9] | 58.7 [53.0 to 64.3]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 61.8 [56.2 to 67.4] | 56.0 [50.5 to 61.6] | 55.8 [50.2 to 61.4]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 62.0 [56.3 to 67.6] | 55.9 [50.3 to 61.5] | 57.2 [51.6 to 62.8]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 58.0 [52.1 to 63.9] | 56.7 [51.1 to 62.2] | 56.3 [50.7 to 61.9]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 61.1 [55.4 to 66.8] | 58.7 [53.1 to 64.3] | 57.1 [51.4 to 62.8]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 60.7 [55.1 to 66.4] | 55.9 [50.3 to 61.5] | 56.2 [50.4 to 62.0]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 58.5 [52.7 to 64.4] | 53.7 [48.1 to 59.4] | 57.0 [51.0 to 63.0]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 59.7 [53.8 to 65.5] | 54.5 [48.9 to 60.1] | 51.5 [45.6 to 57.4]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 60.2 [54.5 to 66.0] | 54.1 [48.3 to 60.0] | 60.7 [54.8 to 66.5]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 59.2 [53.1 to 62.5] | 55.6 [49.8 to 61.4] | 56.6 [50.7 to 62.5]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 58.7 [52.9 to 64.6] | 52.5 [46.7 to 58.3] | 57.0 [51.0 to 62.9]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 59.6 [53.6 to 65.6] | 55.0 [49.2 to 60.7] | 56.5 [50.4 to 62.5]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 56.2 [50.3 to 62.1] | 53.3 [47.5 to 59.1] | 55.8 [49.8 to 61.8]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 58.3 [52.4 to 64.1] | 53.5 [47.6 to 59.5] | 57.0 [51.0 to 63.0]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 59.5 [53.6 to 65.4] | 55.0 [49.2 to 60.8] | 58.5 [52.5 to 64.5]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 65.4 [59.5 to 71.2] | 58.0 [52.1 to 63.8] | 58.8 [52.6 to 64.9]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 63.7 [58.0 to 69.3] | 54.0 [48.2 to 59.9] | 65.3 [59.5 to 71.2]

8. Secondary Outcome: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 57.8 [52.3 to 63.2] | 61.8 [56.4 to 67.2] | 59.2 [53.7 to 64.6]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 67.0 [61.9 to 72.2] | 68.8 [63.7 to 73.9] | 66.0 [60.7 to 71.2]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 70.9 [65.9 to 76.0] | 74.3 [69.4 to 79.2] | 72.5 [67.4 to 77.5]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 75.4 [70.6 to 80.2] | 74.6 [69.9 to 79.4] | 69.6 [64.4 to 74.8]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 76.0 [71.2 to 80.8] | 79.5 [75.1 to 84.0] | 71.4 [66.3 to 76.6]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 78.3 [73.7 to 83.0] | 76.3 [71.6 to 80.9] | 72.2 [67.2 to 77.2]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 76.8 [72.0 to 81.7] | 79.4 [74.8 to 83.9] | 77.2 [72.4 to 81.9]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 80.0 [75.4 to 84.6] | 78.3 [73.6 to 83.0] | 75.9 [70.9 to 80.8]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 79.0 [74.2 to 83.8] | 80.0 [75.4 to 84.6] | 78.4 [73.7 to 83.2]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 79.5 [74.8 to 84.2] | 78.0 [73.2 to 82.7] | 79.8 [75.1 to 84.5]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 84.0 [79.7 to 88.3] | 77.5 [72.8 to 82.3] | 81.9 [77.5 to 86.3]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 81.3 [76.7 to 86.0] | 81.5 [77.1 to 85.9] | 77.2 [72.4 to 82.0]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 81.7 [77.1 to 86.3] | 78.2 [73.5 to 83.0] | 77.1 [72.2 to 82.0]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 78.6 [73.8 to 83.4] | 79.2 [74.5 to 83.8] | 80.3 [75.7 to 84.9]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 75.7 [70.5 to 80.8] | 75.9 [71.0 to 80.9] | 80.3 [75.4 to 85.1]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 77.6 [72.6 to 82.6] | 77.3 [72.5 to 82.0] | 72.5 [67.2 to 77.8]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 77.0 [72.0 to 82.1] | 76.0 [70.9 to 81.0] | 78.5 [73.5 to 83.4]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 79.5 [74.5 to 84.4] | 76.7 [71.6 to 81.7] | 76.1 [70.8 to 81.3]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 75.6 [70.5 to 80.8] | 73.8 [68.7 to 78.9] | 72.6 [67.1 to 78.0]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 74.9 [69.7 to 80.2] | 75.4 [70.3 to 80.5] | 77.4 [72.2 to 82.5]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 73.1 [67.7 to 78.4] | 79.9 [75.2 to 84.7] | 75.2 [70.0 to 80.3]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 74.2 [69.0 to 79.5] | 74.3 [69.2 to 79.5] | 77.5 [72.4 to 82.6]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 76.5 [71.3 to 81.7] | 76.6 [71.6 to 81.6] | 77.4 [72.2 to 82.6]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 80.9 [76.1 to 85.7] | 76.2 [71.2 to 81.2] | 76.0 [70.7 to 81.3]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 80.0 [75.1 to 84.8] | 75.3 [70.3 to 80.4] | 81.3 [76.3 to 86.2]

9. Secondary Outcome: Percentage of Participants Gaining ≥0 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 85.1 [81.2 to 89.0] | 89.2 [85.8 to 92.7] | 89.3 [85.9 to 92.8]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 90.2 [86.9 to 93.5] | 91.3 [88.2 to 94.4] | 90.3 [87.0 to 93.6]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 90.8 [87.6 to 94.0] | 92.7 [89.8 to 95.6] | 90.4 [87.1 to 93.7]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 92.4 [89.4 to 95.3] | 91.1 [88.0 to 94.3] | 90.9 [87.7 to 94.1]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 92.2 [89.1 to 95.3] | 91.7 [88.6 to 94.8] | 93.9 [91.2 to 96.6]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 91.5 [88.3 to 94.7] | 91.5 [88.5 to 94.6] | 91.5 [88.4 to 94.7]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 92.2 [89.1 to 95.4] | 94.3 [91.7 to 96.8] | 94.0 [91.4 to 96.7]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 91.4 [88.2 to 94.7] | 90.9 [87.6 to 94.2] | 92.8 [89.8 to 95.8]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 92.4 [89.3 to 95.5] | 90.5 [87.1 to 93.8] | 95.0 [92.5 to 97.5]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 92.0 [88.8 to 95.2] | 92.3 [89.3 to 95.4] | 93.1 [90.1 to 96.0]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 91.8 [88.5 to 95.1] | 91.2 [88.0 to 94.5] | 92.6 [89.6 to 95.6]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 93.7 [90.7 to 96.7] | 91.0 [87.7 to 94.3] | 91.4 [88.2 to 94.6]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 93.6 [90.7 to 96.5] | 90.4 [86.9 to 93.8] | 91.9 [88.7 to 95.1]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 92.7 [89.6 to 95.7] | 91.5 [88.3 to 94.7] | 90.9 [87.5 to 94.3]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 89.3 [85.6 to 93.0] | 88.5 [84.9 to 92.2] | 92.6 [89.5 to 95.8]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 91.3 [87.9 to 94.6] | 89.7 [86.2 to 93.2] | 87.4 [83.4 to 91.4]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 89.4 [85.6 to 93.2] | 90.5 [87.0 to 94.0] | 91.3 [87.8 to 94.7]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 89.1 [85.2 to 93.0] | 90.4 [86.8 to 94.0] | 88.4 [84.5 to 92.3]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 89.6 [86.0 to 93.3] | 86.3 [82.3 to 90.3] | 90.3 [86.7 to 94.0]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 86.6 [82.5 to 90.8] | 88.5 [84.7 to 92.3] | 88.6 [84.6 to 92.5]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 87.1 [83.0 to 91.2] | 90.2 [86.7 to 93.7] | 87.9 [83.9 to 91.9]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 84.4 [80.0 to 88.9] | 89.5 [85.9 to 93.1] | 88.1 [84.1 to 92.0]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 86.7 [82.5 to 90.9] | 86.7 [82.6 to 90.7] | 87.1 [82.9 to 91.3]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 86.5 [82.3 to 90.7] | 87.0 [83.0 to 91.0] | 89.1 [85.2 to 93.1]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 86.1 [81.8 to 90.3] | 87.5 [83.7 to 91.4] | 91.1 [87.5 to 94.7]

10. Secondary Outcome: Percentage of Participants Gaining ≥15, ≥10, ≥5, or ≥0 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, Treatment-Naive Population
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. Only participants with at least one non-missing, valid assessment at Weeks 48, 52, or 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 208 | 231 | 213
Percentage of participants
  Gaining ≥15 Letters | 32.9 [26.7 to 39.0] | 29.4 [23.9 to 34.9] | 32.7 [26.5 to 38.8]
  Gaining ≥10 Letters | 58.3 [51.8 to 64.8] | 55.5 [49.3 to 61.7] | 56.1 [49.6 to 62.5]
  Gaining ≥5 Letters | 81.8 [76.5 to 87.0] | 79.6 [74.5 to 84.7] | 80.6 [75.4 to 85.8]
  Gaining ≥0 Letters | 93.2 [89.8 to 96.7] | 92.2 [88.8 to 95.6] | 92.0 [88.4 to 95.6]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.2, 95% CI 2-sided [-8.5 to 8.9]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = -3.5, 95% CI 2-sided [-11.8 to 4.8]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 2.2, 95% CI 2-sided [-6.9 to 11.4]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = -0.8, 95% CI 2-sided [-9.8 to 8.1]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 5]; Test type: Other; Difference in CMH Weighted Percentage = 1.2, 95% CI 2-sided [-6.2 to 8.5]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 6]; Test type: Other; Difference in CMH Weighted Percentage = -1.1, 95% CI 2-sided [-8.3 to 6.2]
Statistical Analysis 7: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 7]; Test type: Other; Difference in CMH Weighted Percentage = 1.2, 95% CI 2-sided [-3.8 to 6.2]
Statistical Analysis 8: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 5, analysis 8]; Test type: Other; Difference in CMH Weighted Percentage = 0.2, 95% CI 2-sided [-4.8 to 5.2]

11. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: Treatment-Naive (TN) Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization, grouped according to the treatment assigned at randomization. At each timepoint, only participants with non-missing, valid assessments were included in the analysis. One participant in Arm B: Faricimab 6 mg PTI was excluded from the TN Population for the final analysis due to a late report of prior anti-VEGF treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 13.9 [9.7 to 18.0] | 10.7 [7.0 to 14.4] | 10.3 [6.6 to 14.1]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 14.7 [10.3 to 19.1] | 17.9 [13.2 to 22.5] | 15.7 [11.2 to 20.1]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 19.9 [15.0 to 24.8] | 23.2 [18.1 to 28.3] | 19.7 [14.8 to 24.6]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 23.3 [18.0 to 28.5] | 26.0 [20.8 to 31.2] | 23.5 [18.2 to 28.7]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 25.9 [20.4 to 31.4] | 22.7 [17.5 to 27.9] | 22.0 [16.9 to 27.1]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 30.2 [24.4 to 35.9] | 24.5 [19.2 to 29.7] | 24.3 [18.9 to 29.6]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 29.8 [23.9 to 35.6] | 28.3 [22.7 to 33.8] | 26.5 [20.8 to 32.1]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 34.4 [28.4 to 40.5] | 27.9 [22.1 to 33.6] | 25.1 [19.6 to 30.7]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 34.1 [28.0 to 40.2] | 34.2 [28.3 to 40.1] | 28.9 [23.2 to 34.5]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 37.8 [31.4 to 44.1] | 32.5 [26.6 to 38.4] | 28.4 [22.6 to 34.2]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 36.1 [29.9 to 42.3] | 30.4 [24.6 to 36.2] | 35.0 [28.7 to 41.2]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 32.8 [26.4 to 39.2] | 31.2 [25.5 to 36.9] | 31.7 [25.7 to 37.8]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 34.1 [27.9 to 40.3] | 32.7 [26.9 to 38.6] | 33.9 [27.7 to 40.2]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 39.2 [33.0 to 45.5] | 30.6 [24.8 to 36.3] | 37.6 [31.1 to 44.2]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 37.4 [31.0 to 43.7] | 32.5 [26.5 to 38.4] | 36.2 [29.9 to 42.5]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 39.8 [33.5 to 46.1] | 31.1 [25.2 to 37.0] | 31.9 [25.8 to 38.0]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 36.0 [29.7 to 42.3] | 33.4 [27.2 to 39.7] | 36.4 [30.0 to 42.8]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 35.1 [28.5 to 41.6] | 33.7 [27.5 to 39.9] | 34.7 [28.2 to 41.2]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 37.2 [30.9 to 43.6] | 32.5 [26.4 to 38.6] | 34.5 [28.0 to 40.9]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 40.1 [33.5 to 46.8] | 33.8 [27.6 to 40.0] | 37.0 [30.5 to 43.6]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 40.1 [33.6 to 46.6] | 32.0 [25.9 to 38.1] | 39.4 [32.8 to 45.9]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 39.5 [32.9 to 46.1] | 29.9 [23.8 to 35.9] | 38.4 [31.8 to 45.0]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 42.8 [36.1 to 49.6] | 38.0 [31.7 to 44.2] | 42.5 [35.6 to 49.4]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 42.9 [36.1 to 49.7] | 35.9 [29.8 to 41.9] | 35.9 [29.2 to 42.5]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 43.9 [37.1 to 50.8] | 33.0 [26.9 to 39.0] | 40.9 [34.0 to 47.9]

12. Secondary Outcome: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 29.4 [23.9 to 34.9] | 28.9 [23.3 to 34.5] | 26.9 [21.3 to 32.4]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 38.2 [32.3 to 44.1] | 42.2 [36.1 to 48.3] | 33.1 [27.2 to 38.9]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 45.2 [39.0 to 51.4] | 46.9 [40.7 to 53.1] | 43.9 [37.7 to 50.1]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 52.3 [46.2 to 58.5] | 51.4 [45.4 to 57.4] | 41.7 [35.5 to 48.0]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 53.4 [47.2 to 59.6] | 51.1 [44.9 to 57.4] | 45.5 [39.2 to 51.8]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 57.8 [51.6 to 64.1] | 53.1 [46.9 to 59.2] | 49.3 [43.1 to 55.5]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 59.7 [53.4 to 66.1] | 53.1 [46.9 to 59.4] | 55.3 [49.0 to 61.6]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 61.2 [54.7 to 67.6] | 50.6 [44.2 to 57.1] | 55.7 [49.2 to 62.1]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 58.8 [52.3 to 65.2] | 57.8 [51.5 to 64.0] | 59.6 [53.1 to 66.0]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 61.3 [55.0 to 67.7] | 56.8 [50.6 to 63.1] | 58.5 [52.2 to 64.9]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 61.6 [55.0 to 68.2] | 56.8 [50.5 to 63.1] | 61.1 [54.7 to 67.4]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 57.4 [50.6 to 64.2] | 58.0 [51.7 to 64.2] | 58.1 [51.7 to 64.6]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 60.9 [54.4 to 67.4] | 61.6 [55.3 to 67.8] | 60.0 [53.5 to 66.5]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 61.0 [54.6 to 67.4] | 58.6 [52.3 to 64.9] | 58.6 [51.9 to 65.3]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 57.9 [51.3 to 64.5] | 57.1 [50.8 to 63.5] | 56.2 [49.5 to 63.0]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 58.4 [51.8 to 65.0] | 56.2 [49.9 to 62.5] | 53.7 [46.9 to 60.4]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 58.9 [52.4 to 65.4] | 54.4 [47.8 to 61.0] | 60.7 [54.0 to 67.3]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 58.4 [51.5 to 65.4] | 57.5 [51.0 to 64.1] | 59.3 [52.5 to 66.0]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 58.2 [51.5 to 64.9] | 54.0 [47.5 to 60.6] | 57.5 [50.8 to 64.3]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 60.4 [53.6 to 67.2] | 58.1 [51.6 to 64.6] | 57.0 [50.2 to 63.9]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 55.9 [49.1 to 62.8] | 56.5 [50.0 to 63.1] | 57.1 [50.3 to 63.8]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 57.1 [50.3 to 63.9] | 53.6 [46.9 to 60.3] | 58.8 [52.0 to 65.6]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 58.8 [51.9 to 65.6] | 57.0 [50.4 to 63.5] | 60.5 [53.7 to 67.2]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 64.7 [58.0 to 71.4] | 58.4 [51.9 to 65.0] | 59.8 [52.9 to 66.7]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 63.0 [56.5 to 69.5] | 55.2 [48.7 to 61.7] | 66.2 [59.5 to 72.8]

13. Secondary Outcome: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 57.9 [51.8 to 64.1] | 62.2 [56.1 to 68.3] | 58.3 [52.1 to 64.5]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 65.6 [59.7 to 71.4] | 68.3 [62.5 to 74.1] | 65.3 [59.3 to 71.2]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 71.1 [65.4 to 76.8] | 74.7 [69.2 to 80.2] | 72.4 [66.7 to 78.1]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 76.4 [71.1 to 81.7] | 75.5 [70.1 to 80.8] | 69.1 [63.2 to 75.1]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 76.5 [71.1 to 81.9] | 80.4 [75.4 to 85.3] | 72.5 [66.8 to 78.3]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 78.0 [72.7 to 83.3] | 77.4 [72.2 to 82.6] | 72.2 [66.5 to 77.9]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 77.2 [71.7 to 82.7] | 79.7 [74.6 to 84.9] | 76.9 [71.5 to 82.3]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 81.1 [75.9 to 86.3] | 80.0 [74.8 to 85.3] | 77.1 [71.6 to 82.6]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 77.4 [71.8 to 83.0] | 81.4 [76.2 to 86.5] | 79.3 [73.9 to 84.7]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 78.6 [73.1 to 84.0] | 79.7 [74.4 to 85.0] | 81.5 [76.2 to 86.7]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 83.7 [78.7 to 88.6] | 79.3 [74.0 to 84.5] | 85.8 [81.1 to 90.5]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 79.9 [74.4 to 85.4] | 84.0 [79.2 to 88.7] | 79.0 [73.6 to 84.4]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 81.8 [76.6 to 87.0] | 80.3 [75.1 to 85.4] | 79.4 [73.9 to 84.8]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 78.2 [72.7 to 83.7] | 78.7 [73.4 to 84.0] | 82.4 [77.2 to 87.7]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 75.1 [69.4 to 80.9] | 77.3 [71.8 to 82.8] | 80.3 [74.8 to 85.7]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 76.3 [70.5 to 82.1] | 79.0 [73.7 to 84.2] | 73.0 [66.9 to 79.0]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 75.4 [69.6 to 81.3] | 77.6 [72.0 to 83.2] | 78.2 [72.6 to 83.9]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 78.4 [72.8 to 84.1] | 77.7 [72.1 to 83.4] | 77.3 [71.5 to 83.1]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 75.6 [69.7 to 81.5] | 76.1 [70.4 to 81.7] | 73.6 [67.5 to 79.8]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 75.2 [69.3 to 81.1] | 78.2 [72.6 to 83.8] | 78.5 [72.7 to 84.2]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 72.3 [66.1 to 78.5] | 80.5 [75.2 to 85.9] | 76.3 [70.5 to 82.2]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 73.9 [67.8 to 80.0] | 75.9 [70.2 to 81.7] | 80.6 [75.1 to 86.2]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 73.7 [67.6 to 79.9] | 77.4 [71.8 to 83.0] | 80.2 [74.5 to 85.9]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 78.7 [73.0 to 84.4] | 77.5 [72.0 to 83.0] | 76.9 [70.9 to 82.8]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 79.0 [73.4 to 84.6] | 78.2 [72.7 to 83.7] | 81.7 [76.2 to 87.3]

14. Secondary Outcome: Percentage of Participants Gaining ≥0 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 84.9 [80.5 to 89.3] | 88.5 [84.5 to 92.5] | 88.8 [84.9 to 92.8]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 89.3 [85.4 to 93.1] | 90.6 [87.0 to 94.2] | 90.1 [86.3 to 93.9]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 90.1 [86.4 to 93.9] | 92.9 [89.7 to 96.1] | 90.6 [86.9 to 94.3]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 91.3 [87.7 to 94.8] | 90.9 [87.3 to 94.5] | 91.3 [87.7 to 94.9]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 91.9 [88.4 to 95.4] | 92.9 [89.6 to 96.1] | 93.9 [90.9 to 97.0]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 90.9 [87.3 to 94.6] | 92.6 [89.3 to 95.9] | 92.2 [88.7 to 95.7]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 91.9 [88.4 to 95.5] | 95.2 [92.5 to 98.0] | 94.5 [91.6 to 97.5]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 91.2 [87.4 to 95.0] | 90.5 [86.6 to 94.4] | 93.5 [90.2 to 96.8]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 91.5 [87.8 to 95.3] | 90.5 [86.7 to 94.4] | 96.2 [93.7 to 98.8]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 91.6 [87.9 to 95.3] | 92.8 [89.5 to 96.2] | 94.8 [91.9 to 97.8]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 91.8 [88.1 to 95.6] | 91.5 [87.8 to 95.1] | 95.3 [92.4 to 98.1]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 93.5 [90.0 to 96.9] | 91.1 [87.5 to 94.8] | 92.9 [89.4 to 96.4]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 94.3 [91.1 to 97.4] | 91.0 [87.3 to 94.8] | 93.3 [89.9 to 96.7]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 93.9 [90.7 to 97.1] | 92.4 [89.0 to 95.9] | 91.0 [87.1 to 95.0]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 88.5 [84.2 to 92.8] | 87.8 [83.4 to 92.1] | 93.0 [89.5 to 96.5]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 90.5 [86.5 to 94.4] | 89.5 [85.5 to 93.5] | 88.5 [84.1 to 92.9]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 89.6 [85.4 to 93.8] | 90.7 [86.8 to 94.6] | 90.5 [86.4 to 94.5]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 89.1 [84.7 to 93.5] | 89.7 [85.6 to 93.9] | 87.7 [83.1 to 92.3]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 89.6 [85.5 to 93.8] | 88.5 [84.2 to 92.7] | 89.7 [85.4 to 94.0]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 86.4 [81.5 to 91.2] | 89.7 [85.6 to 93.8] | 88.9 [84.4 to 93.3]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 87.6 [83.0 to 92.2] | 91.1 [87.3 to 94.9] | 88.0 [83.5 to 92.5]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 84.7 [79.7 to 89.7] | 90.2 [86.2 to 94.1] | 90.6 [86.4 to 94.7]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 85.5 [80.6 to 90.5] | 86.3 [81.7 to 90.9] | 88.9 [84.3 to 93.4]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 84.8 [79.8 to 89.9] | 87.8 [83.4 to 92.2] | 89.3 [84.9 to 93.7]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 85.3 [80.4 to 90.3] | 89.0 [84.9 to 93.1] | 91.8 [87.8 to 95.7]

15. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 268 | 293 | 279
Percentage of participants
  Avoiding a Loss of ≥15 Letters | 98.9 [97.6 to 100.0] | 98.7 [97.4 to 100.0] | 98.6 [97.2 to 99.9]
  Avoiding a Loss of ≥10 Letters | 98.1 [96.5 to 99.7] | 98.0 [96.4 to 99.6] | 98.2 [96.7 to 99.7]
  Avoiding a Loss of ≥5 Letters | 96.7 [94.5 to 98.8] | 97.0 [95.0 to 98.9] | 95.4 [93.0 to 97.8]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥15 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.3, 95% CI 2-sided [-1.6 to 2.1]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥15 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-1.8 to 1.9]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥10 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.1, 95% CI 2-sided [-2.3 to 2.1]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥10 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = -0.3, 95% CI 2-sided [-2.4 to 1.9]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥5 letters in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 1.3, 95% CI 2-sided [-1.9 to 4.5]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants avoiding a loss of ≥5 letters in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W; Test type: Other; Difference in CMH Weighted Percentage = 1.6, 95% CI 2-sided [-1.5 to 4.6]

16. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The weighted estimates of the percentage of participants avoiding a loss of letters in BCVA from baseline were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 99.4 [98.5 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 99.7 [99.1 to 100.0] | 100.0 [100.0 to 100.0] | 99.7 [99.1 to 100.0]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 99.7 [99.0 to 100.0] | 99.7 [99.1 to 100.0] | 99.7 [99.1 to 100.0]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 99.7 [99.0 to 100.0]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 99.6 [99.0 to 100.0] | 99.3 [98.4 to 100.0] | 99.3 [98.4 to 100.0]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 99.3 [98.4 to 100.0] | 99.3 [98.4 to 100.0] | 99.3 [98.4 to 100.0]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 99.7 [99.0 to 100.0] | 99.3 [98.4 to 100.0] | 99.0 [97.8 to 100.0]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 98.9 [97.7 to 100.0] | 98.9 [97.8 to 100.0] | 98.5 [97.2 to 99.9]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 99.3 [98.3 to 100.0] | 99.0 [97.9 to 100.0] | 98.9 [97.8 to 100.0]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 98.9 [97.6 to 100.0] | 98.6 [97.3 to 99.9] | 99.3 [98.3 to 100.0]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 99.6 [98.8 to 100.0] | 99.0 [97.8 to 100.0] | 98.5 [97.2 to 99.9]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 99.6 [98.8 to 100.0] | 98.3 [96.8 to 99.8] | 99.3 [98.3 to 100.0]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 98.4 [96.9 to 99.9] | 98.9 [97.8 to 100.0] | 99.6 [99.0 to 100.0]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 98.5 [97.0 to 100.0] | 99.3 [98.4 to 100.0] | 98.9 [97.6 to 100.0]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 98.8 [97.5 to 100.0] | 98.9 [97.7 to 100.0] | 98.0 [96.4 to 99.7]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 98.4 [96.9 to 99.9] | 98.3 [96.8 to 99.8] | 96.9 [94.8 to 99.0]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 98.4 [96.9 to 99.9] | 98.2 [96.6 to 99.8] | 97.6 [95.8 to 99.5]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 98.9 [97.6 to 100.0] | 98.8 [97.6 to 100.0] | 97.6 [95.8 to 99.5]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 96.9 [94.8 to 99.0] | 98.2 [96.6 to 99.8] | 97.6 [95.7 to 99.5]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 96.4 [94.1 to 98.7] | 98.1 [96.5 to 99.7] | 97.5 [95.6 to 99.5]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 96.2 [93.9 to 98.5] | 99.3 [98.3 to 100.0] | 97.3 [95.3 to 99.3]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 94.9 [92.2 to 97.6] | 98.1 [96.5 to 99.7] | 97.6 [95.7 to 99.5]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 96.0 [93.6 to 98.4] | 97.4 [95.5 to 99.3] | 97.1 [95.0 to 99.2]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 95.5 [92.9 to 98.1] | 97.8 [96.0 to 99.5] | 98.4 [96.8 to 99.9]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 96.1 [93.7 to 98.4] | 96.3 [94.1 to 98.5] | 96.1 [93.7 to 98.5]

17. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 16
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 99.4 [98.5 to 100.0] | 99.3 [98.4 to 100.0] | 99.4 [98.5 to 100.0]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 99.0 [98.0 to 100.0] | 99.4 [98.5 to 100.0] | 99.0 [98.0 to 100.0]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 98.7 [97.5 to 99.9] | 99.0 [98.0 to 100.0] | 99.3 [98.5 to 100.0]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 99.7 [99.0 to 100.0] | 99.7 [99.0 to 100.0] | 99.3 [98.4 to 100.0]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 98.6 [97.3 to 99.9] | 99.0 [97.9 to 100.0] | 99.0 [97.9 to 100.0]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 98.2 [96.7 to 99.8] | 99.3 [98.4 to 100.0] | 98.7 [97.4 to 99.9]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 99.7 [99.0 to 100.0] | 99.0 [97.8 to 100.0] | 99.0 [97.8 to 100.0]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 98.5 [97.1 to 99.9] | 98.6 [97.3 to 99.9] | 97.5 [95.7 to 99.2]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 98.9 [97.7 to 100.0] | 98.7 [97.4 to 99.9] | 98.2 [96.7 to 99.8]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 98.1 [96.5 to 99.7] | 97.9 [96.3 to 99.6] | 98.6 [97.2 to 99.9]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 98.5 [97.0 to 100.0] | 98.6 [97.3 to 100.0] | 98.2 [96.6 to 99.7]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 98.4 [96.8 to 99.9] | 96.5 [94.5 to 98.6] | 98.9 [97.8 to 100.0]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 97.7 [95.9 to 99.5] | 98.2 [96.7 to 99.8] | 98.6 [97.2 to 99.9]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 98.5 [97.0 to 100.0] | 98.6 [97.2 to 99.9] | 97.0 [95.0 to 99.0]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 98.0 [96.3 to 99.7] | 97.1 [95.2 to 99.1] | 96.5 [94.3 to 98.7]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 97.7 [95.9 to 99.5] | 97.3 [95.4 to 99.1] | 96.5 [94.3 to 98.7]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 96.4 [94.1 to 98.7] | 96.3 [94.1 to 98.5] | 96.0 [93.6 to 98.4]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 96.4 [94.1 to 98.7] | 98.1 [96.4 to 99.7] | 97.2 [95.2 to 99.2]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 95.7 [93.2 to 98.1] | 97.4 [95.5 to 99.3] | 96.8 [94.6 to 99.0]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 95.2 [92.5 to 97.8] | 96.7 [94.6 to 98.8] | 95.9 [93.4 to 98.3]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 94.6 [91.9 to 97.3] | 98.5 [97.1 to 99.9] | 95.3 [92.7 to 97.9]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 93.3 [90.3 to 96.4] | 97.0 [95.0 to 99.0] | 95.1 [92.4 to 97.7]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 93.6 [90.6 to 96.6] | 94.8 [92.1 to 97.4] | 95.4 [92.9 to 98.0]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 93.4 [90.3 to 96.5] | 95.5 [93.0 to 98.0] | 95.3 [92.7 to 98.0]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 94.8 [92.2 to 97.5] | 94.9 [92.3 to 97.5] | 94.8 [92.0 to 97.6]

18. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, ITT Population
Description: as for outcome 16
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 95.1 [92.8 to 97.5] | 97.4 [95.6 to 99.2] | 97.7 [96.1 to 99.4]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 96.7 [94.7 to 98.7] | 97.1 [95.3 to 98.9] | 97.1 [95.2 to 98.9]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 97.4 [95.6 to 99.2] | 96.7 [94.7 to 98.7] | 97.0 [95.1 to 98.9]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 97.7 [96.0 to 99.4] | 97.7 [96.0 to 99.4] | 96.6 [94.6 to 98.7]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 96.9 [95.0 to 98.9] | 96.7 [94.7 to 98.7] | 97.3 [95.5 to 99.1]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 96.5 [94.4 to 98.6] | 96.4 [94.4 to 98.5] | 96.4 [94.3 to 98.4]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 96.1 [93.9 to 98.4] | 97.3 [95.5 to 99.1] | 97.9 [96.3 to 99.5]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 96.4 [94.3 to 98.6] | 96.5 [94.4 to 98.6] | 95.0 [92.5 to 97.5]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 97.5 [95.7 to 99.3] | 96.6 [94.5 to 98.6] | 97.5 [95.7 to 99.3]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 96.7 [94.6 to 98.8] | 95.9 [93.6 to 98.1] | 96.7 [94.7 to 98.8]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 96.3 [94.0 to 98.5] | 95.8 [93.5 to 98.1] | 96.3 [94.1 to 98.5]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 96.4 [94.2 to 98.7] | 95.2 [92.7 to 97.6] | 96.1 [93.8 to 98.3]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 96.2 [93.9 to 98.4] | 94.7 [92.1 to 97.3] | 96.7 [94.5 to 98.8]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 95.6 [93.1 to 98.0] | 96.8 [94.7 to 98.8] | 96.6 [94.5 to 98.7]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 95.0 [92.3 to 97.6] | 94.6 [92.0 to 97.2] | 95.3 [92.8 to 97.8]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 95.9 [93.5 to 98.2] | 92.8 [89.8 to 95.8] | 93.3 [90.3 to 96.3]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 94.8 [92.1 to 97.6] | 93.7 [90.8 to 96.6] | 94.9 [92.1 to 97.6]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 94.0 [91.0 to 96.9] | 94.6 [91.9 to 97.4] | 92.9 [89.7 to 96.0]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 93.7 [90.8 to 96.7] | 92.3 [89.2 to 95.5] | 94.7 [92.0 to 97.5]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 92.4 [89.1 to 95.7] | 93.8 [90.9 to 96.6] | 93.4 [90.4 to 96.4]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 92.7 [89.6 to 95.8] | 93.3 [90.3 to 96.2] | 92.9 [89.9 to 96.0]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 89.9 [86.2 to 93.5] | 91.7 [88.5 to 95.0] | 93.4 [90.4 to 96.5]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 91.7 [88.3 to 95.1] | 90.7 [87.3 to 94.2] | 92.9 [89.7 to 96.1]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 90.1 [86.4 to 93.8] | 91.1 [87.7 to 94.5] | 92.8 [89.5 to 96.1]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 91.6 [88.2 to 95.0] | 90.4 [87.0 to 93.9] | 93.6 [90.5 to 96.7]

19. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters in BCVA From Baseline in the Study Eye Averaged Over Weeks 48, 52, and 56, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 208 | 231 | 213
Percentage of participants
  Avoiding a Loss of ≥15 Letters | 98.5 [96.9 to 100.0] | 98.7 [97.2 to 100.0] | 98.6 [97.0 to 100.0]
  Avoiding a Loss of ≥10 Letters | 98.1 [96.2 to 99.9] | 97.8 [96.0 to 99.7] | 98.1 [96.3 to 99.9]
  Avoiding a Loss of ≥5 Letters | 97.6 [95.5 to 99.7] | 97.4 [95.4 to 99.4] | 96.2 [93.7 to 98.8]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-2.3 to 2.2]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 0.1, 95% CI 2-sided [-2.0 to 2.2]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [-2.7 to 2.6]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = -0.3, 95% CI 2-sided [-2.9 to 2.3]
Statistical Analysis 5: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 5]; Test type: Other; Difference in CMH Weighted Percentage = 1.3, 95% CI 2-sided [-2.0 to 4.7]
Statistical Analysis 6: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 15, analysis 6]; Test type: Other; Difference in CMH Weighted Percentage = 1.2, 95% CI 2-sided [-2.1 to 4.4]

20. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The weighted estimates of the percentage of participants avoiding a loss of letters in BCVA from baseline were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 99.6 [98.8 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 99.6 [98.8 to 100.0]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 100.0 [100.0 to 100.0] | 99.6 [98.8 to 100.0] | 99.6 [98.8 to 100.0]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 99.6 [98.7 to 100.0]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 100.0 [100.0 to 100.0] | 99.2 [98.0 to 100.0] | 99.6 [98.7 to 100.0]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 99.2 [98.0 to 100.0] | 99.2 [98.0 to 100.0] | 99.6 [98.8 to 100.0]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 99.6 [98.8 to 100.0] | 99.6 [98.7 to 100.0] | 99.1 [97.9 to 100.0]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 98.6 [97.1 to 100.0] | 99.1 [97.8 to 100.0] | 99.1 [97.8 to 100.0]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 99.0 [97.7 to 100.0] | 99.2 [98.1 to 100.0] | 99.1 [97.8 to 100.0]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 99.0 [97.7 to 100.0] | 99.1 [97.9 to 100.0] | 99.5 [98.6 to 100.0]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 99.5 [98.5 to 100.0] | 99.1 [97.9 to 100.0] | 99.1 [97.8 to 100.0]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 99.5 [98.5 to 100.0] | 98.3 [96.6 to 99.9] | 99.5 [98.6 to 100.0]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 99.0 [97.6 to 100.0] | 98.6 [97.1 to 100.0] | 100.0 [100.0 to 100.0]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 98.1 [96.2 to 99.9] | 99.1 [97.9 to 100.0] | 98.5 [96.9 to 100.0]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 99.0 [97.7 to 100.0] | 98.6 [97.1 to 100.0] | 98.5 [96.8 to 100.0]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 99.0 [97.7 to 100.0] | 98.2 [96.5 to 99.9] | 97.0 [94.7 to 99.4]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 99.0 [97.6 to 100.0] | 97.7 [95.7 to 99.7] | 97.5 [95.4 to 99.7]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 99.5 [98.5 to 100.0] | 98.5 [96.9 to 100.0] | 97.5 [95.3 to 99.7]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 97.5 [95.3 to 99.7] | 97.7 [95.7 to 99.7] | 97.5 [95.3 to 99.6]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 96.8 [94.3 to 99.3] | 98.1 [96.3 to 99.9] | 97.9 [95.8 to 99.9]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 96.9 [94.5 to 99.3] | 99.1 [97.9 to 100.0] | 97.0 [94.7 to 99.4]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 94.9 [91.8 to 98.0] | 98.1 [96.3 to 99.9] | 97.4 [95.2 to 99.6]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 96.4 [93.7 to 99.0] | 97.2 [94.9 to 99.4] | 97.4 [95.1 to 99.6]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 95.3 [92.3 to 98.3] | 97.7 [95.7 to 99.7] | 98.5 [96.8 to 100.0]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 95.5 [92.6 to 98.4] | 96.3 [93.7 to 98.8] | 96.7 [94.1 to 99.3]

21. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 20
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 99.6 [98.8 to 100.0] | 99.2 [98.0 to 100.0] | 99.2 [98.0 to 100.0]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 99.2 [98.0 to 100.0] | 99.2 [98.1 to 100.0] | 98.8 [97.4 to 100.0]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 99.2 [98.1 to 100.0] | 99.2 [98.1 to 100.0] | 99.2 [98.0 to 100.0]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 99.6 [98.8 to 100.0] | 99.6 [98.8 to 100.0] | 99.1 [97.9 to 100.0]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 98.7 [97.3 to 100.0] | 98.8 [97.3 to 100.0] | 99.1 [97.9 to 100.0]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 97.8 [95.9 to 99.7] | 99.2 [98.0 to 100.0] | 99.6 [98.8 to 100.0]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 99.6 [98.8 to 100.0] | 99.1 [97.9 to 100.0] | 99.1 [97.9 to 100.0]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 98.2 [96.4 to 99.9] | 99.1 [97.8 to 100.0] | 98.6 [97.0 to 100.0]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 98.6 [97.0 to 100.0] | 98.7 [97.3 to 100.0] | 98.6 [97.0 to 100.0]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 98.5 [96.9 to 100.0] | 98.7 [97.2 to 100.0] | 98.6 [97.1 to 100.0]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 98.1 [96.2 to 99.9] | 98.7 [97.2 to 100.0] | 98.6 [97.0 to 100.0]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 99.0 [97.5 to 100.0] | 96.5 [94.1 to 98.9] | 99.5 [98.6 to 100.0]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 98.5 [96.9 to 100.0] | 97.8 [95.8 to 99.7] | 99.0 [97.7 to 100.0]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 98.1 [96.2 to 99.9] | 98.7 [97.2 to 100.0] | 96.6 [94.1 to 99.1]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 98.5 [96.9 to 100.0] | 96.4 [93.9 to 98.8] | 97.0 [94.6 to 99.4]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 98.6 [96.9 to 100.0] | 96.9 [94.7 to 99.2] | 97.0 [94.7 to 99.4]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 97.0 [94.6 to 99.4] | 95.4 [92.6 to 98.2] | 95.5 [92.6 to 98.4]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 97.9 [95.8 to 99.9] | 98.1 [96.2 to 99.9] | 97.5 [95.3 to 99.7]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 96.0 [93.2 to 98.7] | 97.2 [95.0 to 99.4] | 96.4 [93.8 to 99.0]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 95.8 [92.9 to 98.6] | 96.3 [93.7 to 98.8] | 96.3 [93.6 to 99.0]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 95.9 [93.1 to 98.7] | 98.6 [97.1 to 100.0] | 95.5 [92.6 to 98.4]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 93.9 [90.5 to 97.2] | 96.7 [94.4 to 99.1] | 95.3 [92.3 to 98.3]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 93.8 [90.4 to 97.2] | 94.8 [91.8 to 97.8] | 95.8 [93.0 to 98.6]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 92.7 [89.0 to 96.4] | 96.2 [93.6 to 98.8] | 95.7 [92.9 to 98.6]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 94.5 [91.3 to 97.6] | 94.5 [91.4 to 97.5] | 96.1 [93.3 to 98.9]

22. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 20
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 95.5 [92.9 to 98.1] | 97.1 [95.0 to 99.2] | 97.5 [95.6 to 99.5]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 96.3 [93.9 to 98.6] | 97.1 [95.1 to 99.2] | 96.3 [93.9 to 98.7]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 97.5 [95.6 to 99.5] | 97.1 [95.0 to 99.2] | 97.0 [94.9 to 99.2]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 97.1 [95.0 to 99.2] | 98.3 [96.7 to 99.9] | 97.0 [94.7 to 99.2]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 96.6 [94.3 to 98.9] | 96.2 [93.8 to 98.6] | 97.8 [96.0 to 99.7]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 96.1 [93.6 to 98.6] | 97.1 [95.1 to 99.2] | 97.4 [95.4 to 99.5]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 96.8 [94.5 to 99.1] | 97.8 [96.0 to 99.7] | 98.2 [96.4 to 99.9]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 96.8 [94.5 to 99.1] | 96.4 [93.9 to 98.8] | 95.8 [93.1 to 98.5]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 97.2 [95.0 to 99.4] | 96.5 [94.1 to 98.9] | 98.1 [96.3 to 99.9]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 96.7 [94.3 to 99.1] | 96.9 [94.7 to 99.1] | 97.2 [95.0 to 99.4]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 96.2 [93.6 to 98.8] | 96.0 [93.4 to 98.5] | 97.7 [95.6 to 99.7]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 96.4 [93.9 to 99.0] | 95.6 [93.0 to 98.3] | 96.2 [93.7 to 98.8]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 97.5 [95.4 to 99.7] | 94.6 [91.7 to 97.6] | 98.0 [96.2 to 99.9]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 96.7 [94.2 to 99.1] | 97.8 [95.8 to 99.7] | 96.6 [94.1 to 99.1]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 95.7 [92.9 to 98.4] | 94.1 [91.1 to 97.2] | 95.5 [92.6 to 98.4]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 96.2 [93.7 to 98.8] | 92.1 [88.6 to 95.6] | 94.1 [90.8 to 97.3]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 95.0 [92.0 to 98.0] | 93.0 [89.6 to 96.4] | 94.0 [90.7 to 97.3]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 94.8 [91.7 to 97.9] | 94.2 [90.9 to 97.4] | 92.4 [88.7 to 96.1]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 94.0 [90.7 to 97.3] | 93.2 [89.9 to 96.5] | 93.8 [90.4 to 97.2]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 92.7 [89.0 to 96.4] | 94.5 [91.4 to 97.5] | 94.1 [90.8 to 97.5]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 93.8 [90.4 to 97.2] | 93.9 [90.7 to 97.1] | 93.5 [90.0 to 96.9]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 90.8 [86.7 to 94.8] | 92.1 [88.5 to 95.7] | 93.7 [90.2 to 97.1]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 91.3 [87.4 to 95.3] | 90.6 [86.7 to 94.5] | 93.1 [89.4 to 96.7]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 88.5 [84.0 to 93.0] | 92.0 [88.4 to 95.7] | 93.0 [89.4 to 96.7]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 90.4 [86.3 to 94.5] | 91.7 [88.1 to 95.4] | 94.5 [91.2 to 97.8]

23. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: as for outcome 5
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: ITT Population and Treatment-Naive Population. Only participants with at least one non-missing, valid assessment at Weeks 48, 52, or 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 268 | 294 | 279
Percentage of participants
  ITT Population | 38.3 [32.6 to 44.0] | 32.4 [27.2 to 37.6] | 33.5 [28.1 to 38.9]
  Treatment-Naive Population: number analyzed (Participants) | 208 | 232 | 213
  Treatment-Naive Population | 38.1 [31.7 to 44.5] | 34.4 [28.5 to 40.4] | 35.5 [29.2 to 41.9]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W for the ITT Population; Test type: Other; Difference in CMH Weighted Percentage = 4.8, 95% CI 2-sided [-3.1 to 12.7]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W for the ITT Population; Test type: Other; Difference in CMH Weighted Percentage = -1.3, 95% CI 2-sided [-8.8 to 6.2]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W for the Treatment-Naive Population; Test type: Other; Difference in CMH Weighted Percentage = 2.6, 95% CI 2-sided [-6.5 to 11.6]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the difference in percentage of participants in Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W for the Treatment-Naive Population; Test type: Other; Difference in CMH Weighted Percentage = -1.3, 95% CI 2-sided [-10.0 to 7.4]

24. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Over Time, ITT Population
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 308 | 309
  Week 4 | 14.7 [11.0 to 18.5] | 13.0 [9.4 to 16.7] | 13.2 [9.5 to 16.9]
  Week 8: number analyzed (Participants) | 306 | 313 | 309
  Week 8 | 17.3 [13.1 to 21.5] | 20.4 [16.0 to 24.8] | 18.1 [13.8 to 22.3]
  Week 12: number analyzed (Participants) | 306 | 305 | 302
  Week 12 | 23.2 [18.5 to 27.8] | 25.5 [20.8 to 30.3] | 22.7 [18.1 to 27.3]
  Week 16: number analyzed (Participants) | 301 | 306 | 296
  Week 16 | 27.3 [22.4 to 32.2] | 28.0 [23.2 to 32.8] | 25.8 [21.0 to 30.7]
  Week 20: number analyzed (Participants) | 294 | 304 | 295
  Week 20 | 28.7 [23.7 to 33.8] | 24.0 [19.3 to 28.8] | 26.5 [21.7 to 31.4]
  Week 24: number analyzed (Participants) | 294 | 307 | 297
  Week 24 | 33.3 [28.0 to 38.6] | 29.1 [24.0 to 34.1] | 27.6 [22.6 to 32.6]
  Week 28: number analyzed (Participants) | 285 | 295 | 287
  Week 28 | 34.9 [29.4 to 40.3] | 30.7 [25.6 to 35.8] | 28.8 [23.6 to 34.0]
  Week 32: number analyzed (Participants) | 278 | 284 | 280
  Week 32 | 39.0 [33.5 to 44.6] | 30.4 [25.2 to 35.7] | 27.5 [22.4 to 32.6]
  Week 36: number analyzed (Participants) | 275 | 282 | 275
  Week 36 | 36.3 [30.9 to 41.8] | 35.8 [30.4 to 41.2] | 33.2 [27.9 to 38.5]
  Week 40: number analyzed (Participants) | 276 | 287 | 274
  Week 40 | 41.0 [35.3 to 46.6] | 34.2 [28.9 to 39.5] | 34.5 [29.0 to 40.0]
  Week 44: number analyzed (Participants) | 270 | 287 | 272
  Week 44 | 40.6 [35.0 to 46.3] | 33.5 [28.1 to 38.8] | 38.5 [32.9 to 44.1]
  Week 48: number analyzed (Participants) | 255 | 287 | 278
  Week 48 | 36.6 [30.8 to 42.4] | 32.6 [27.4 to 37.8] | 33.9 [28.4 to 39.3]
  Week 52: number analyzed (Participants) | 268 | 282 | 271
  Week 52 | 39.3 [33.7 to 45.0] | 34.7 [29.3 to 40.2] | 38.4 [32.7 to 44.1]
  Week 56: number analyzed (Participants) | 268 | 284 | 261
  Week 56 | 43.4 [37.7 to 49.2] | 33.2 [27.9 to 38.5] | 40.3 [34.4 to 46.2]
  Week 60: number analyzed (Participants) | 262 | 277 | 255
  Week 60 | 41.2 [35.3 to 47.0] | 34.2 [28.8 to 39.6] | 39.0 [33.2 to 44.8]
  Week 64: number analyzed (Participants) | 258 | 291 | 259
  Week 64 | 44.4 [38.5 to 50.2] | 31.6 [26.4 to 36.8] | 35.0 [29.4 to 40.7]
  Week 68: number analyzed (Participants) | 255 | 273 | 255
  Week 68 | 40.2 [34.4 to 46.0] | 33.5 [27.9 to 39.0] | 39.0 [33.2 to 44.8]
  Week 72: number analyzed (Participants) | 246 | 262 | 250
  Week 72 | 41.0 [35.0 to 47.1] | 34.4 [28.8 to 39.9] | 36.1 [30.4 to 41.8]
  Week 76: number analyzed (Participants) | 257 | 274 | 251
  Week 76 | 39.7 [34.0 to 45.5] | 35.7 [30.2 to 41.3] | 39.1 [33.2 to 44.9]
  Week 80: number analyzed (Participants) | 248 | 270 | 250
  Week 80 | 43.4 [37.4 to 49.4] | 32.8 [27.4 to 38.2] | 38.7 [32.7 to 44.6]
  Week 84: number analyzed (Participants) | 253 | 266 | 255
  Week 84 | 41.7 [35.9 to 47.5] | 33.8 [28.2 to 39.4] | 40.5 [34.7 to 46.4]
  Week 88: number analyzed (Participants) | 255 | 268 | 247
  Week 88 | 42.6 [36.8 to 48.4] | 32.5 [27.0 to 38.0] | 41.7 [35.7 to 47.6]
  Week 92: number analyzed (Participants) | 250 | 269 | 242
  Week 92 | 45.6 [39.7 to 51.6] | 38.3 [32.7 to 43.9] | 45.0 [38.9 to 51.2]
  Week 96: number analyzed (Participants) | 245 | 268 | 241
  Week 96 | 46.0 [39.9 to 52.1] | 37.2 [31.7 to 42.7] | 40.6 [34.5 to 46.7]
  Week 100: number analyzed (Participants) | 252 | 272 | 237
  Week 100 | 44.5 [38.4 to 50.5] | 34.3 [28.8 to 39.7] | 44.3 [38.1 to 50.5]

25. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 245 | 242
  Week 4 | 15.1 [10.8 to 19.3] | 13.5 [9.4 to 17.6] | 12.8 [8.6 to 17.0]
  Week 8: number analyzed (Participants) | 245 | 248 | 242
  Week 8 | 17.0 [12.4 to 21.7] | 22.2 [17.0 to 27.3] | 17.7 [13.0 to 22.4]
  Week 12: number analyzed (Participants) | 243 | 243 | 236
  Week 12 | 22.6 [17.4 to 27.8] | 26.3 [21.0 to 31.6] | 22.7 [17.6 to 27.9]
  Week 16: number analyzed (Participants) | 242 | 243 | 230
  Week 16 | 26.1 [20.6 to 31.5] | 30.0 [24.4 to 35.5] | 26.1 [20.6 to 31.6]
  Week 20: number analyzed (Participants) | 233 | 241 | 230
  Week 20 | 28.4 [22.7 to 34.1] | 26.2 [20.7 to 31.7] | 25.9 [20.5 to 31.4]
  Week 24: number analyzed (Participants) | 232 | 243 | 232
  Week 24 | 34.2 [28.2 to 40.3] | 30.5 [24.8 to 36.3] | 27.3 [21.7 to 32.9]
  Week 28: number analyzed (Participants) | 224 | 232 | 222
  Week 28 | 35.4 [29.1 to 41.6] | 32.9 [27.0 to 38.9] | 29.6 [23.7 to 35.6]
  Week 32: number analyzed (Participants) | 217 | 220 | 216
  Week 32 | 38.4 [32.0 to 44.7] | 31.5 [25.5 to 37.5] | 28.9 [23.0 to 34.8]
  Week 36: number analyzed (Participants) | 212 | 221 | 209
  Week 36 | 37.0 [30.7 to 43.3] | 38.0 [31.9 to 44.2] | 34.6 [28.5 to 40.8]
  Week 40: number analyzed (Participants) | 214 | 223 | 211
  Week 40 | 41.4 [34.9 to 47.8] | 36.4 [30.2 to 42.5] | 34.6 [28.3 to 40.9]
  Week 44: number analyzed (Participants) | 209 | 224 | 211
  Week 44 | 40.3 [33.8 to 46.7] | 34.3 [28.2 to 40.4] | 40.7 [34.2 to 47.2]
  Week 48: number analyzed (Participants) | 199 | 225 | 212
  Week 48 | 36.7 [30.1 to 43.4] | 34.9 [28.9 to 40.9] | 36.5 [30.1 to 42.9]
  Week 52: number analyzed (Participants) | 210 | 224 | 207
  Week 52 | 39.1 [32.6 to 45.6] | 37.0 [30.8 to 43.2] | 39.8 [33.2 to 46.4]
  Week 56: number analyzed (Participants) | 210 | 225 | 200
  Week 56 | 44.7 [38.1 to 51.2] | 35.2 [29.1 to 41.3] | 41.7 [35.0 to 48.5]
  Week 60: number analyzed (Participants) | 209 | 219 | 200
  Week 60 | 40.9 [34.3 to 47.5] | 36.9 [30.6 to 43.2] | 39.2 [32.7 to 45.8]
  Week 64: number analyzed (Participants) | 205 | 229 | 203
  Week 64 | 44.0 [37.4 to 50.6] | 33.6 [27.5 to 39.7] | 35.4 [29.0 to 41.8]
  Week 68: number analyzed (Participants) | 202 | 215 | 200
  Week 68 | 39.7 [33.2 to 46.2] | 35.5 [29.1 to 41.9] | 40.0 [33.4 to 46.6]
  Week 72: number analyzed (Participants) | 192 | 206 | 196
  Week 72 | 40.0 [33.1 to 46.8] | 37.7 [31.2 to 44.2] | 38.3 [31.7 to 45.0]
  Week 76: number analyzed (Participants) | 199 | 217 | 195
  Week 76 | 40.6 [34.0 to 47.2] | 37.8 [31.4 to 44.2] | 39.1 [32.4 to 45.8]
  Week 80: number analyzed (Participants) | 190 | 211 | 193
  Week 80 | 44.9 [38.0 to 51.8] | 37.3 [30.9 to 43.7] | 40.9 [34.1 to 47.6]
  Week 84: number analyzed (Participants) | 194 | 210 | 199
  Week 84 | 43.1 [36.5 to 49.8] | 36.0 [29.6 to 42.4] | 41.4 [34.8 to 48.1]
  Week 88: number analyzed (Participants) | 195 | 212 | 191
  Week 88 | 42.3 [35.6 to 49.1] | 33.5 [27.2 to 39.8] | 41.5 [34.7 to 48.2]
  Week 92: number analyzed (Participants) | 193 | 210 | 188
  Week 92 | 47.1 [40.2 to 54.0] | 42.6 [36.1 to 49.2] | 45.2 [38.2 to 52.1]
  Week 96: number analyzed (Participants) | 191 | 211 | 189
  Week 96 | 44.6 [37.7 to 51.5] | 39.5 [33.1 to 45.8] | 41.4 [34.4 to 48.3]
  Week 100: number analyzed (Participants) | 197 | 214 | 183
  Week 100 | 45.6 [38.7 to 52.5] | 36.9 [30.6 to 43.2] | 44.9 [37.8 to 52.0]

26. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥69 vs. <69 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 268 | 293 | 279
Percentage of participants
  ITT Population | 73.2 [68.2 to 78.3] | 71.6 [66.7 to 76.4] | 68.5 [63.6 to 73.5]
  Treatment-Naive Population: number analyzed (Participants) | 208 | 231 | 213
  Treatment-Naive Population | 73.6 [68.0 to 79.3] | 74.2 [68.9 to 79.5] | 72.1 [66.6 to 77.7]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 4.7, 95% CI 2-sided [-2.4 to 11.8]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 2.8, 95% CI 2-sided [-4.1 to 9.8]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 1.5, 95% CI 2-sided [-6.5 to 9.4]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 1.7, 95% CI 2-sided [-6.0 to 9.3]

27. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥69 vs. <69 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 306 | 309
  Week 4 | 56.7 [51.6 to 61.7] | 57.8 [53.2 to 62.4] | 54.4 [49.7 to 59.1]
  Week 8: number analyzed (Participants) | 305 | 311 | 309
  Week 8 | 61.3 [56.4 to 66.2] | 65.7 [61.1 to 70.3] | 59.4 [54.7 to 64.1]
  Week 12: number analyzed (Participants) | 305 | 303 | 302
  Week 12 | 68.0 [63.2 to 72.8] | 67.8 [63.2 to 72.4] | 65.2 [60.4 to 70.0]
  Week 16: number analyzed (Participants) | 300 | 304 | 296
  Week 16 | 66.8 [61.9 to 71.7] | 69.2 [64.6 to 73.7] | 64.6 [59.7 to 69.6]
  Week 20: number analyzed (Participants) | 294 | 302 | 295
  Week 20 | 69.6 [64.8 to 74.5] | 67.3 [62.5 to 72.0] | 66.0 [61.2 to 70.7]
  Week 24: number analyzed (Participants) | 293 | 306 | 297
  Week 24 | 70.6 [65.7 to 75.6] | 69.1 [64.4 to 73.8] | 65.5 [60.6 to 70.4]
  Week 28: number analyzed (Participants) | 284 | 295 | 287
  Week 28 | 72.0 [67.1 to 76.9] | 69.9 [65.2 to 74.5] | 67.0 [62.2 to 71.9]
  Week 32: number analyzed (Participants) | 277 | 284 | 280
  Week 32 | 72.6 [67.6 to 77.7] | 71.9 [67.1 to 76.7] | 67.3 [62.4 to 72.2]
  Week 36: number analyzed (Participants) | 275 | 281 | 275
  Week 36 | 71.4 [66.3 to 76.4] | 69.6 [64.6 to 74.5] | 70.1 [65.2 to 75.1]
  Week 40: number analyzed (Participants) | 275 | 286 | 274
  Week 40 | 73.8 [68.9 to 78.6] | 70.8 [65.9 to 75.6] | 70.4 [65.4 to 75.4]
  Week 44: number analyzed (Participants) | 269 | 286 | 272
  Week 44 | 73.7 [68.7 to 78.8] | 71.1 [66.3 to 75.9] | 69.0 [64.0 to 73.9]
  Week 48: number analyzed (Participants) | 255 | 286 | 278
  Week 48 | 73.1 [67.8 to 78.3] | 73.0 [68.1 to 77.9] | 67.1 [62.1 to 72.0]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 74.5 [69.5 to 79.5] | 69.8 [64.8 to 74.8] | 71.0 [66.1 to 75.9]
  Week 56: number analyzed (Participants) | 267 | 283 | 261
  Week 56 | 74.7 [69.7 to 79.8] | 73.4 [68.6 to 78.2] | 71.9 [66.8 to 76.9]
  Week 60: number analyzed (Participants) | 261 | 277 | 255
  Week 60 | 70.3 [64.9 to 75.7] | 67.1 [62.0 to 72.3] | 69.4 [64.3 to 74.5]
  Week 64: number analyzed (Participants) | 258 | 290 | 259
  Week 64 | 74.5 [69.5 to 79.6] | 68.1 [63.0 to 73.2] | 68.2 [63.0 to 73.5]
  Week 68: number analyzed (Participants) | 254 | 272 | 255
  Week 68 | 71.9 [66.6 to 77.2] | 68.4 [63.2 to 73.6] | 72.3 [67.2 to 77.4]
  Week 72: number analyzed (Participants) | 245 | 261 | 250
  Week 72 | 68.8 [63.2 to 74.3] | 72.2 [67.2 to 77.3] | 66.2 [60.8 to 71.6]
  Week 76: number analyzed (Participants) | 257 | 273 | 251
  Week 76 | 70.1 [64.8 to 75.5] | 69.0 [63.9 to 74.2] | 70.7 [65.3 to 76.1]
  Week 80: number analyzed (Participants) | 247 | 269 | 250
  Week 80 | 72.4 [67.0 to 77.8] | 70.9 [65.8 to 76.0] | 69.5 [64.0 to 74.9]
  Week 84: number analyzed (Participants) | 253 | 265 | 255
  Week 84 | 72.7 [67.4 to 78.0] | 71.6 [66.5 to 76.8] | 71.4 [66.0 to 76.7]
  Week 88: number analyzed (Participants) | 254 | 267 | 247
  Week 88 | 68.7 [63.3 to 74.2] | 70.3 [65.1 to 75.5] | 71.3 [65.9 to 76.6]
  Week 92: number analyzed (Participants) | 249 | 269 | 242
  Week 92 | 71.6 [66.1 to 77.0] | 73.5 [68.4 to 78.6] | 69.5 [64.0 to 74.9]
  Week 96: number analyzed (Participants) | 244 | 267 | 241
  Week 96 | 74.9 [69.5 to 80.3] | 73.1 [68.0 to 78.2] | 73.2 [67.9 to 78.5]
  Week 100: number analyzed (Participants) | 251 | 271 | 237
  Week 100 | 73.5 [68.1 to 78.9] | 70.0 [64.8 to 75.1] | 76.4 [71.2 to 81.6]

28. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥69 vs. <69 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 243 | 242
  Week 4 | 57.5 [51.9 to 63.1] | 59.9 [54.8 to 64.9] | 56.0 [50.7 to 61.4]
  Week 8: number analyzed (Participants) | 244 | 246 | 242
  Week 8 | 62.3 [56.8 to 67.7] | 67.0 [61.9 to 72.1] | 59.9 [54.5 to 65.2]
  Week 12: number analyzed (Participants) | 242 | 241 | 236
  Week 12 | 68.9 [63.6 to 74.1] | 70.2 [65.1 to 75.3] | 67.5 [62.1 to 73.0]
  Week 16: number analyzed (Participants) | 241 | 241 | 230
  Week 16 | 66.8 [61.3 to 72.3] | 70.7 [65.7 to 75.7] | 65.0 [59.4 to 70.6]
  Week 20: number analyzed (Participants) | 233 | 239 | 230
  Week 20 | 70.2 [64.7 to 75.6] | 69.2 [64.0 to 74.3] | 67.4 [62.1 to 72.8]
  Week 24: number analyzed (Participants) | 231 | 242 | 232
  Week 24 | 71.1 [65.6 to 76.5] | 71.7 [66.6 to 76.8] | 66.2 [60.8 to 71.7]
  Week 28: number analyzed (Participants) | 223 | 232 | 222
  Week 28 | 73.5 [68.1 to 79.0] | 71.0 [65.9 to 76.1] | 69.4 [64.0 to 74.8]
  Week 32: number analyzed (Participants) | 216 | 220 | 216
  Week 32 | 74.3 [68.7 to 80.0] | 74.8 [69.4 to 80.1] | 70.2 [64.6 to 75.8]
  Week 36: number analyzed (Participants) | 212 | 220 | 209
  Week 36 | 71.8 [66.0 to 77.5] | 71.2 [65.6 to 76.8] | 72.4 [66.9 to 77.9]
  Week 40: number analyzed (Participants) | 213 | 222 | 211
  Week 40 | 74.0 [68.6 to 79.5] | 73.7 [68.4 to 79.0] | 72.3 [66.7 to 77.9]
  Week 44: number analyzed (Participants) | 208 | 223 | 211
  Week 44 | 73.8 [68.1 to 79.4] | 74.3 [69.1 to 79.6] | 73.5 [68.0 to 78.9]
  Week 48: number analyzed (Participants) | 199 | 224 | 212
  Week 48 | 73.1 [67.3 to 79.0] | 76.2 [70.9 to 81.5] | 70.5 [65.0 to 75.9]
  Week 52: number analyzed (Participants) | 209 | 223 | 207
  Week 52 | 73.9 [68.2 to 79.5] | 73.3 [67.7 to 78.8] | 75.5 [70.1 to 80.9]
  Week 56: number analyzed (Participants) | 209 | 224 | 200
  Week 56 | 75.9 [70.3 to 81.5] | 75.5 [70.3 to 80.7] | 74.7 [69.1 to 80.3]
  Week 60: number analyzed (Participants) | 208 | 219 | 200
  Week 60 | 69.9 [63.9 to 76.0] | 70.9 [65.2 to 76.7] | 71.5 [65.8 to 77.2]
  Week 64: number analyzed (Participants) | 205 | 228 | 203
  Week 64 | 73.7 [67.9 to 79.4] | 70.6 [65.0 to 76.2] | 70.4 [64.5 to 76.2]
  Week 68: number analyzed (Participants) | 201 | 214 | 200
  Week 68 | 71.8 [65.8 to 77.7] | 68.4 [62.5 to 74.3] | 73.9 [68.2 to 79.5]
  Week 72: number analyzed (Participants) | 191 | 205 | 196
  Week 72 | 67.0 [60.6 to 73.3] | 73.9 [68.2 to 79.6] | 68.6 [62.6 to 74.6]
  Week 76: number analyzed (Participants) | 199 | 216 | 195
  Week 76 | 70.3 [64.1 to 76.4] | 72.1 [66.4 to 77.8] | 71.7 [65.7 to 77.8]
  Week 80: number analyzed (Participants) | 189 | 210 | 193
  Week 80 | 73.2 [67.0 to 79.3] | 72.5 [66.8 to 78.3] | 72.6 [66.6 to 78.6]
  Week 84: number analyzed (Participants) | 194 | 209 | 199
  Week 84 | 73.4 [67.4 to 79.4] | 72.2 [66.4 to 78.0] | 72.5 [66.6 to 78.5]
  Week 88: number analyzed (Participants) | 194 | 211 | 191
  Week 88 | 68.1 [62.0 to 74.3] | 70.4 [64.5 to 76.2] | 75.3 [69.3 to 81.2]
  Week 92: number analyzed (Participants) | 192 | 210 | 188
  Week 92 | 70.5 [64.2 to 76.8] | 74.5 [68.6 to 80.4] | 73.2 [67.2 to 79.2]
  Week 96: number analyzed (Participants) | 190 | 210 | 189
  Week 96 | 72.7 [66.4 to 79.0] | 74.8 [69.1 to 80.5] | 73.8 [67.9 to 79.8]
  Week 100: number analyzed (Participants) | 196 | 213 | 183
  Week 100 | 71.2 [64.9 to 77.4] | 70.7 [64.8 to 76.6] | 77.7 [71.9 to 83.5]

29. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: as for outcome 5
Time Frame: Baseline, average of Weeks 48, 52, and 56
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 268 | 294 | 279
Percentage of participants
  ITT Population | 0.8 [0.0 to 1.8] | 0.0 [0.0 to 0.0] | 0.7 [0.0 to 1.7]
  Treatment-Naive Population: number analyzed (Participants) | 208 | 232 | 213
  Treatment-Naive Population | 1.0 [0.0 to 2.3] | 0.0 [0.0 to 0.0] | 0.5 [0.0 to 1.4]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.1, 95% CI 2-sided [-1.4 to 1.5]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = -0.7, 95% CI 2-sided [-1.6 to 0.2]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.5, 95% CI 2-sided [-1.1 to 2.1]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = -0.5, 95% CI 2-sided [-1.4 to 0.4]

30. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Over Time, ITT Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement invisual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 307 | 308 | 309
  Week 4 | 1.6 [0.2 to 3.0] | 1.7 [0.2 to 3.1] | 0.3 [0.0 to 1.0]
  Week 8: number analyzed (Participants) | 306 | 313 | 309
  Week 8 | 1.3 [0.0 to 2.6] | 0.6 [0.0 to 1.5] | 0.3 [0.0 to 1.0]
  Week 12: number analyzed (Participants) | 306 | 305 | 302
  Week 12 | 1.3 [0.1 to 2.6] | 0.7 [0.0 to 1.6] | 0.6 [0.0 to 1.5]
  Week 16: number analyzed (Participants) | 301 | 306 | 296
  Week 16 | 0.3 [0.0 to 1.0] | 0.3 [0.0 to 0.9] | 0.7 [0.0 to 1.5]
  Week 20: number analyzed (Participants) | 294 | 304 | 295
  Week 20 | 1.0 [0.0 to 2.2] | 0.3 [0.0 to 0.9] | 1.0 [0.0 to 2.1]
  Week 24: number analyzed (Participants) | 294 | 307 | 297
  Week 24 | 0.7 [0.0 to 1.7] | 0.3 [0.0 to 1.0] | 1.3 [0.1 to 2.6]
  Week 28: number analyzed (Participants) | 285 | 295 | 287
  Week 28 | 1.1 [0.0 to 2.2] | 0.3 [0.0 to 1.0] | 0.7 [0.0 to 1.6]
  Week 32: number analyzed (Participants) | 278 | 284 | 280
  Week 32 | 0.7 [0.0 to 1.7] | 1.4 [0.1 to 2.8] | 1.1 [0.0 to 2.3]
  Week 36: number analyzed (Participants) | 275 | 282 | 275
  Week 36 | 0.7 [0.0 to 1.7] | 1.3 [0.1 to 2.6] | 0.4 [0.0 to 1.0]
  Week 40: number analyzed (Participants) | 276 | 287 | 274
  Week 40 | 1.1 [0.0 to 2.4] | 1.4 [0.1 to 2.7] | 1.1 [0.0 to 2.3]
  Week 44: number analyzed (Participants) | 270 | 287 | 272
  Week 44 | 0.4 [0.0 to 1.1] | 1.0 [0.0 to 2.2] | 1.1 [0.0 to 2.3]
  Week 48: number analyzed (Participants) | 255 | 287 | 278
  Week 48 | 0.8 [0.0 to 1.9] | 0.7 [0.0 to 1.6] | 1.4 [0.1 to 2.7]
  Week 52: number analyzed (Participants) | 268 | 282 | 271
  Week 52 | 0.4 [0.0 to 1.2] | 0.4 [0.0 to 1.1] | 1.1 [0.0 to 2.2]
  Week 56: number analyzed (Participants) | 268 | 284 | 261
  Week 56 | 1.1 [0.0 to 2.4] | 1.0 [0.0 to 2.2] | 0.8 [0.0 to 1.8]
  Week 60: number analyzed (Participants) | 262 | 277 | 255
  Week 60 | 1.2 [0.0 to 2.5] | 0.7 [0.0 to 1.7] | 1.5 [0.1 to 2.9]
  Week 64: number analyzed (Participants) | 258 | 291 | 259
  Week 64 | 1.2 [0.0 to 2.4] | 0.7 [0.0 to 1.6] | 2.0 [0.3 to 3.7]
  Week 68: number analyzed (Participants) | 255 | 273 | 255
  Week 68 | 1.2 [0.0 to 2.5] | 1.1 [0.0 to 2.4] | 0.4 [0.0 to 1.1]
  Week 72: number analyzed (Participants) | 246 | 262 | 250
  Week 72 | 1.2 [0.0 to 2.5] | 1.9 [0.3 to 3.6] | 1.5 [0.1 to 3.0]
  Week 76: number analyzed (Participants) | 257 | 274 | 251
  Week 76 | 2.7 [0.8 to 4.7] | 1.8 [0.2 to 3.4] | 2.0 [0.3 to 3.7]
  Week 80: number analyzed (Participants) | 248 | 270 | 250
  Week 80 | 2.4 [0.6 to 4.3] | 2.6 [0.7 to 4.6] | 1.6 [0.1 to 3.1]
  Week 84: number analyzed (Participants) | 253 | 266 | 255
  Week 84 | 2.7 [0.7 to 4.6] | 1.2 [0.0 to 2.5] | 1.9 [0.3 to 3.5]
  Week 88: number analyzed (Participants) | 255 | 268 | 247
  Week 88 | 2.3 [0.5 to 4.1] | 1.9 [0.3 to 3.4] | 1.2 [0.0 to 2.5]
  Week 92: number analyzed (Participants) | 250 | 269 | 242
  Week 92 | 3.2 [1.0 to 5.4] | 0.8 [0.0 to 1.8] | 1.6 [0.1 to 3.1]
  Week 96: number analyzed (Participants) | 245 | 268 | 241
  Week 96 | 2.9 [0.8 to 5.0] | 2.3 [0.5 to 4.1] | 2.0 [0.3 to 3.7]
  Week 100: number analyzed (Participants) | 252 | 272 | 237
  Week 100 | 2.7 [0.7 to 4.7] | 3.3 [1.2 to 5.5] | 2.5 [0.5 to 4.4]

31. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Over Time, Treatment-Naive Population
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 4: number analyzed (Participants) | 245 | 245 | 242
  Week 4 | 2.0 [0.3 to 3.8] | 1.7 [0.1 to 3.2] | 0.4 [0.0 to 1.2]
  Week 8: number analyzed (Participants) | 245 | 248 | 242
  Week 8 | 1.6 [0.1 to 3.2] | 0.8 [0.0 to 1.9] | 0.4 [0.0 to 1.2]
  Week 12: number analyzed (Participants) | 243 | 243 | 236
  Week 12 | 1.2 [0.0 to 2.6] | 0.4 [0.0 to 1.2] | 0.8 [0.0 to 2.0]
  Week 16: number analyzed (Participants) | 242 | 243 | 230
  Week 16 | 0.4 [0.0 to 1.2] | 0.4 [0.0 to 1.2] | 0.9 [0.0 to 2.0]
  Week 20: number analyzed (Participants) | 233 | 241 | 230
  Week 20 | 0.9 [0.0 to 2.1] | 0.4 [0.0 to 1.2] | 0.9 [0.0 to 2.0]
  Week 24: number analyzed (Participants) | 232 | 243 | 232
  Week 24 | 0.9 [0.0 to 2.1] | 0.4 [0.0 to 1.2] | 0.8 [0.0 to 2.0]
  Week 28: number analyzed (Participants) | 224 | 232 | 222
  Week 28 | 1.3 [0.0 to 2.8] | 0.4 [0.0 to 1.3] | 0.4 [0.0 to 1.3]
  Week 32: number analyzed (Participants) | 217 | 220 | 216
  Week 32 | 0.9 [0.0 to 2.2] | 1.4 [0.0 to 2.9] | 0.5 [0.0 to 1.4]
  Week 36: number analyzed (Participants) | 212 | 221 | 209
  Week 36 | 1.0 [0.0 to 2.3] | 1.7 [0.1 to 3.4] | 0.5 [0.0 to 1.4]
  Week 40: number analyzed (Participants) | 214 | 223 | 211
  Week 40 | 1.0 [0.0 to 2.2] | 1.8 [0.1 to 3.5] | 0.5 [0.0 to 1.4]
  Week 44: number analyzed (Participants) | 209 | 224 | 211
  Week 44 | 0.5 [0.0 to 1.4] | 1.3 [0.0 to 2.8] | 0.5 [0.0 to 1.4]
  Week 48: number analyzed (Participants) | 199 | 225 | 212
  Week 48 | 1.0 [0.0 to 2.4] | 0.9 [0.0 to 2.1] | 0.5 [0.0 to 1.4]
  Week 52: number analyzed (Participants) | 210 | 224 | 207
  Week 52 | 0.0 [0.0 to 0.0] | 0.5 [0.0 to 1.4] | 0.0 [0.0 to 0.0]
  Week 56: number analyzed (Participants) | 210 | 225 | 200
  Week 56 | 1.4 [0.0 to 3.0] | 0.9 [0.0 to 2.0] | 1.0 [0.0 to 2.4]
  Week 60: number analyzed (Participants) | 209 | 219 | 200
  Week 60 | 0.9 [0.0 to 2.2] | 0.9 [0.0 to 2.2] | 1.0 [0.0 to 2.4]
  Week 64: number analyzed (Participants) | 205 | 229 | 203
  Week 64 | 0.5 [0.0 to 1.4] | 0.9 [0.0 to 2.0] | 2.0 [0.1 to 4.0]
  Week 68: number analyzed (Participants) | 202 | 215 | 200
  Week 68 | 0.5 [0.0 to 1.5] | 1.4 [0.0 to 3.0] | 0.5 [0.0 to 1.4]
  Week 72: number analyzed (Participants) | 192 | 206 | 196
  Week 72 | 1.0 [0.0 to 2.4] | 1.4 [0.0 to 3.1] | 2.0 [0.1 to 3.9]
  Week 76: number analyzed (Participants) | 199 | 217 | 195
  Week 76 | 2.0 [0.1 to 3.9] | 1.8 [0.1 to 3.6] | 2.6 [0.4 to 4.7]
  Week 80: number analyzed (Participants) | 190 | 211 | 193
  Week 80 | 1.6 [0.0 to 3.4] | 2.9 [0.6 to 5.2] | 1.5 [0.0 to 3.3]
  Week 84: number analyzed (Participants) | 194 | 210 | 199
  Week 84 | 2.1 [0.1 to 4.1] | 1.0 [0.0 to 2.3] | 2.0 [0.1 to 3.9]
  Week 88: number analyzed (Participants) | 195 | 212 | 191
  Week 88 | 1.5 [0.0 to 3.2] | 1.9 [0.1 to 3.7] | 1.6 [0.0 to 3.3]
  Week 92: number analyzed (Participants) | 193 | 210 | 188
  Week 92 | 3.2 [0.7 to 5.6] | 0.5 [0.0 to 1.5] | 2.1 [0.1 to 4.1]
  Week 96: number analyzed (Participants) | 191 | 211 | 189
  Week 96 | 2.7 [0.4 to 5.0] | 2.4 [0.3 to 4.5] | 2.0 [0.1 to 4.0]
  Week 100: number analyzed (Participants) | 197 | 214 | 183
  Week 100 | 3.0 [0.6 to 5.4] | 3.8 [1.2 to 6.3] | 2.1 [0.1 to 4.1]

32. Secondary Outcome: Percentage of Participants With a ≥2-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, ITT Population
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 52, and 96
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and each timepoint were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 16: number analyzed (Participants) | 280 | 289 | 271
  Week 16 | 34.5 [29.1 to 39.8] | 38.0 [32.5 to 43.6] | 34.0 [28.6 to 39.5]
  Week 52: number analyzed (Participants) | 249 | 261 | 246
  Week 52 | 43.4 [37.4 to 49.4] | 43.9 [37.9 to 49.8] | 46.2 [40.2 to 52.2]
  Week 96: number analyzed (Participants) | 214 | 228 | 203
  Week 96 | 53.5 [46.9 to 60.1] | 44.3 [37.9 to 50.7] | 43.8 [37.2 to 50.4]

33. Secondary Outcome: Percentage of Participants With a ≥2-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, Treatment-Naive Population
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy. Ocular imaging assessments were made independently by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters) and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 16: number analyzed (Participants) | 224 | 230 | 209
  Week 16 | 37.2 [31.1 to 43.3] | 39.5 [33.3 to 45.7] | 37.3 [31.0 to 43.7]
  Week 52: number analyzed (Participants) | 195 | 206 | 192
  Week 52 | 46.0 [39.1 to 52.9] | 46.2 [39.4 to 53.1] | 51.3 [44.4 to 58.2]
  Week 96: number analyzed (Participants) | 161 | 177 | 160
  Week 96 | 55.2 [47.6 to 62.8] | 44.1 [36.9 to 51.4] | 48.8 [41.1 to 56.4]

34. Secondary Outcome: Percentage of Participants With a ≥3-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, ITT Population
Description: as for outcome 32
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 16: number analyzed (Participants) | 280 | 289 | 271
  Week 16 | 12.8 [9.0 to 16.7] | 17.0 [12.7 to 21.4] | 13.4 [9.3 to 17.4]
  Week 52: number analyzed (Participants) | 249 | 261 | 246
  Week 52 | 16.3 [11.7 to 20.8] | 19.2 [14.4 to 24.0] | 19.2 [14.4 to 24.0]
  Week 96: number analyzed (Participants) | 214 | 228 | 203
  Week 96 | 25.1 [19.3 to 30.9] | 19.3 [14.2 to 24.5] | 21.8 [16.3 to 27.2]

35. Secondary Outcome: Percentage of Participants With a ≥3-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 33
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 16: number analyzed (Participants) | 224 | 230 | 209
  Week 16 | 14.2 [9.7 to 18.7] | 16.6 [11.8 to 21.4] | 14.4 [9.6 to 19.1]
  Week 52: number analyzed (Participants) | 195 | 206 | 192
  Week 52 | 18.9 [13.4 to 24.4] | 19.0 [13.6 to 24.3] | 21.6 [15.9 to 27.4]
  Week 96: number analyzed (Participants) | 161 | 177 | 160
  Week 96 | 27.9 [21.0 to 34.8] | 19.2 [13.4 to 25.0] | 25.7 [19.0 to 32.4]

36. Secondary Outcome: Percentage of Participants With a ≥4-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, ITT Population
Description: as for outcome 32
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 16: number analyzed (Participants) | 280 | 289 | 271
  Week 16 | 3.6 [1.4 to 5.8] | 8.3 [5.2 to 11.5] | 3.4 [1.2 to 5.5]
  Week 52: number analyzed (Participants) | 249 | 261 | 246
  Week 52 | 4.1 [1.6 to 6.5] | 7.3 [4.1 to 10.4] | 4.9 [2.2 to 7.6]
  Week 96: number analyzed (Participants) | 214 | 228 | 203
  Week 96 | 7.7 [4.1 to 11.2] | 7.3 [4.0 to 10.6] | 5.3 [2.3 to 8.4]

37. Secondary Outcome: Percentage of Participants With a ≥4-Step Diabetic Retinopathy Severity Improvement From Baseline on the ETDRS Diabetic Retinopathy Severity Scale in the Study Eye Over Time, Treatment-Naive Population
Description: as for outcome 33
Time Frame: Baseline, Weeks 16, 52, and 96
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
Percentage of participants
  Week 16: number analyzed (Participants) | 224 | 230 | 209
  Week 16 | 3.6 [1.1 to 6.0] | 6.5 [3.3 to 9.7] | 3.3 [0.9 to 5.8]
  Week 52: number analyzed (Participants) | 195 | 206 | 192
  Week 52 | 5.1 [2.0 to 8.1] | 6.3 [3.0 to 9.7] | 4.6 [1.7 to 7.5]
  Week 96: number analyzed (Participants) | 161 | 177 | 160
  Week 96 | 9.2 [4.8 to 13.7] | 5.6 [2.2 to 9.0] | 6.3 [2.5 to 10.0]

38. Secondary Outcome: Percentage of Participants Without Proliferative Diabetic Retinopathy (PDR) at Baseline Who Developed New PDR at Week 52, ITT and Treatment-Naive Populations
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). PDR was defined as an ETDRS DRSS score of ≥61 on the 7-field/4-wide field color fundus photographs assessment by a central reading center. The weighted percentages of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 215 | 221 | 221
Percentage of participants
  ITT Population | 0.8 [0.0 to 2.0] | 0.9 [0.0 to 2.2] | 0.4 [0.0 to 1.3]
  Treatment-Naive Population: number analyzed (Participants) | 164 | 176 | 171
  Treatment-Naive Population | 0.6 [0.0 to 1.8] | 1.2 [0.0 to 2.8] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-1.0 to 1.8]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 0.5, 95% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.6, 95% CI 2-sided [-0.6 to 1.8]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 1.2, 95% CI 2-sided [-0.4 to 2.8]

39. Secondary Outcome: Percentage of Participants Without High-Risk Proliferative Diabetic Retinopathy (PDR) at Baseline Who Developed High-Risk PDR at Week 52, ITT and Treatment-Naive Populations
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) classifies diabetic retinopathy into 12 severity steps ranging from absence of retinopathy to advanced PDR. High-risk PDR was defined as an ETDRS DRSS score of ≥71 on the 7-field/4-wide field color fundus photographs assessment by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 230 | 250 | 236
Percentage of participants
  ITT Population | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Treatment-Naive Population: number analyzed (Participants) | 178 | 197 | 182
  Treatment-Naive Population | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]

40. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 52, ITT Population
Time Frame: Week 52
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 308
Percentage of participants
  Once Every 4 Weeks | 13.3 [9.5 to 17.1]
  Once Every 8 Weeks | 15.6 [11.5 to 19.6]
  Once Every 12 Weeks | 20.1 [15.6 to 24.6]
  Once Every 16 Weeks | 51.0 [45.4 to 56.6]

41. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 52, Treatment-Naive Population
Time Frame: Week 52
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 245
Percentage of participants
  Once Every 4 Weeks | 11.8 [7.8 to 15.9]
  Once Every 8 Weeks | 13.9 [9.5 to 18.2]
  Once Every 12 Weeks | 20.0 [15.0 to 25.0]
  Once Every 16 Weeks | 54.3 [48.0 to 60.5]

42. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 96, ITT Population
Time Frame: Week 96
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 96.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 287
Percentage of participants
  Once Every 4 Weeks | 10.1 [6.6 to 13.6]
  Once Every 8 Weeks | 11.8 [8.1 to 15.6]
  Once Every 12 Weeks | 13.6 [9.6 to 17.6]
  Once Every 16 Weeks | 64.5 [58.9 to 70.0]

43. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm on a Once Every 4-Weeks, 8-Weeks, 12-Weeks, or 16-Weeks Treatment Interval at Week 96, Treatment-Naive Population
Time Frame: Week 96
Population: Treatment-Naive Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization. Participants were grouped according to the treatment assigned at randomization. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 96.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 227
Percentage of participants
  Once Every 4 Weeks | 9.3 [5.5 to 13.0]
  Once Every 8 Weeks | 9.7 [5.8 to 13.5]
  Once Every 12 Weeks | 12.8 [8.4 to 17.1]
  Once Every 16 Weeks | 68.3 [62.2 to 74.3]

44. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm at Week 52 Who Achieved a Once Every 12-Weeks or 16-Weeks Treatment Interval Without an Interval Decrease Below Once Every 12 Weeks, ITT and Treatment-Naive Populations
Time Frame: From start of PTI (Week 12 or later) until Week 52
Population: ITT Population and Treatment-Naive Population. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 308
Percentage of participants
  ITT Population | 64.3 [58.9 to 69.6]
  Treatment-Naive Population: number analyzed (Participants) | 245
  Treatment-Naive Population | 66.9 [61.0 to 72.8]

45. Secondary Outcome: Percentage of Participants in the Faricimab 6 mg PTI Arm at Week 96 Who Achieved a Once Every 12-Weeks or 16-Weeks Treatment Interval Without an Interval Decrease Below Once Every 12 Weeks, ITT and Treatment-Naive Populations
Time Frame: From start of PTI (Week 12 or later) until Week 96
Population: ITT Population and Treatment-Naive Population. The number analyzed includes all participants in Arm B: Faricimab 6 mg PTI who had not discontinued the study prior to Week 96.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 287
Percentage of participants
  ITT Population | 63.1 [57.5 to 68.7]
  Treatment-Naive Population: number analyzed (Participants) | 227
  Treatment-Naive Population | 65.6 [59.4 to 71.8]

46. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline CST (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment (U.S. and Canada vs. the rest of the world; Asia and rest of the world regions were combined). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: From Baseline through Week 56
Population: ITT Population and Treatment-Naive Population
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
microns
  ITT Population | -195.8 [-204.1 to -187.5] | -187.6 [-195.8 to -179.5] | -170.1 [-178.3 to -161.8]
  Treatment-Naive Population: number analyzed (Participants) | 254 | 254 | 248
  Treatment-Naive Population | -195.0 [-204.2 to -185.9] | -189.4 [-198.3 to -180.4] | -175.1 [-184.2 to -165.9]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Other; Adjusted mean difference = -25.7, 95% CI 2-sided [-37.4 to -14.0], Standard Error of Mean 5.95
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the ITT Population; Test type: Other; Adjusted mean difference = -17.6, 95% CI 2-sided [-29.2 to -6.0], Standard Error of Mean 5.88
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm A: Faricimab 6 mg Q8W minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Other; Adjusted mean difference = -20.0, 95% CI 2-sided [-32.9 to -7.0], Standard Error of Mean 6.59
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; This is the adjusted mean difference for Arm B: Faricimab 6 mg PTI minus Arm C: Aflibercept 2 mg Q8W in the Treatment-Naive Population; Test type: Other; Adjusted mean difference = -14.3, 95% CI 2-sided [-27.1 to -1.5], Standard Error of Mean 6.51

47. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Over Time, ITT Population
Description: as for outcome 46
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
microns
  Week 4 | -106.1 [-115.7 to -96.6] | -113.9 [-123.4 to -104.4] | -107.3 [-116.8 to -97.7]
  Week 8 | -132.0 [-140.9 to -123.0] | -139.6 [-148.4 to -130.8] | -129.6 [-138.5 to -120.6]
  Week 12 | -146.0 [-154.8 to -137.2] | -155.0 [-163.7 to -146.3] | -143.1 [-151.9 to -134.2]
  Week 16 | -162.2 [-170.4 to -154.0] | -167.1 [-175.2 to -158.9] | -151.4 [-159.7 to -143.2]
  Week 20 | -166.8 [-176.0 to -157.6] | -157.2 [-166.3 to -148.1] | -154.6 [-163.8 to -145.4]
  Week 24 | -179.9 [-188.4 to -171.3] | -181.4 [-189.8 to -173.0] | -146.6 [-155.1 to -138.1]
  Week 28 | -164.8 [-173.2 to -156.5] | -184.0 [-192.3 to -175.8] | -165.0 [-173.3 to -156.6]
  Week 32 | -181.9 [-191.4 to -172.4] | -169.4 [-178.9 to -160.0] | -154.8 [-164.3 to -145.3]
  Week 36 | -170.9 [-179.8 to -162.1] | -189.2 [-197.9 to -180.5] | -168.6 [-177.4 to -159.7]
  Week 40 | -191.6 [-200.9 to -182.3] | -183.8 [-193.0 to -174.6] | -160.0 [-169.3 to -150.7]
  Week 44 | -181.7 [-191.0 to -172.3] | -185.9 [-195.1 to -176.7] | -172.3 [-181.7 to -162.9]
  Week 48 | -195.6 [-205.0 to -186.2] | -184.9 [-194.1 to -175.8] | -162.7 [-172.0 to -153.4]
  Week 52 | -188.6 [-197.9 to -179.3] | -186.1 [-195.3 to -177.0] | -176.6 [-185.9 to -167.3]
  Week 56 | -199.0 [-208.4 to -189.7] | -188.5 [-197.7 to -179.4] | -168.2 [-177.5 to -158.8]
  Week 60 | -194.1 [-204.1 to -184.0] | -186.1 [-195.9 to -176.3] | -179.0 [-189.1 to -168.9]
  Week 64 | -197.2 [-206.7 to -187.8] | -189.8 [-199.0 to -180.7] | -172.1 [-181.5 to -162.8]
  Week 68 | -196.2 [-205.2 to -187.1] | -190.3 [-199.2 to -181.5] | -181.4 [-190.4 to -172.4]
  Week 72 | -202.8 [-212.3 to -193.4] | -191.9 [-201.2 to -182.6] | -172.5 [-181.9 to -163.0]
  Week 76 | -198.8 [-207.4 to -190.3] | -191.3 [-199.6 to -182.9] | -185.4 [-194.0 to -176.8]
  Week 80 | -204.0 [-213.4 to -194.6] | -189.7 [-198.8 to -180.5] | -176.7 [-186.1 to -167.3]
  Week 84 | -198.2 [-207.6 to -188.9] | -197.9 [-207.1 to -188.8] | -185.5 [-194.7 to -176.2]
  Week 88 | -201.5 [-211.3 to -191.7] | -194.9 [-204.4 to -185.3] | -177.1 [-186.9 to -167.3]
  Week 92 | -200.5 [-210.2 to -190.9] | -195.4 [-204.7 to -186.1] | -184.0 [-193.7 to -174.4]
  Week 96 | -206.3 [-215.7 to -196.8] | -199.0 [-208.2 to -189.7] | -180.0 [-189.5 to -170.5]
  Week 100 | -201.1 [-210.5 to -191.8] | -196.9 [-206.0 to -187.8] | -192.8 [-202.2 to -183.3]

48. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Over Time, Treatment-Naive Population
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline CST (continuous), baseline BCVA (<64 vs. ≥64 letters), and region of enrollment (U.S. and Canada vs. the rest of the world; Asia and rest of the world regions were combined). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: Treatment-Naive (TN) Population: all participants randomized in the study who had not received any intravitreal anti-VEGF agents in the study eye prior to randomization, grouped according to the treatment assigned at randomization. One participant in Arm B: Faricimab 6 mg PTI was excluded from the TN Population for the final analysis due to a late report of prior anti-VEGF treatment.
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 254 | 254 | 248
microns
  Week 4 | -106.3 [-116.9 to -95.6] | -112.9 [-123.5 to -102.3] | -106.3 [-117.0 to -95.6]
  Week 8 | -131.8 [-141.6 to -122.0] | -140.6 [-150.3 to -130.9] | -130.4 [-140.2 to -120.5]
  Week 12 | -148.8 [-158.4 to -139.2] | -156.6 [-166.2 to -147.1] | -145.3 [-154.9 to -135.6]
  Week 16 | -163.0 [-171.9 to -154.0] | -168.8 [-177.7 to -159.9] | -157.0 [-166.0 to -148.0]
  Week 20 | -170.5 [-180.1 to -160.9] | -162.3 [-171.9 to -152.8] | -160.6 [-170.2 to -150.9]
  Week 24 | -182.4 [-191.5 to -173.3] | -182.9 [-191.9 to -173.9] | -154.6 [-163.8 to -145.5]
  Week 28 | -166.8 [-175.9 to -157.8] | -183.9 [-192.9 to -174.9] | -174.2 [-183.2 to -165.1]
  Week 32 | -183.7 [-194.0 to -173.4] | -168.0 [-178.2 to -157.7] | -161.0 [-171.4 to -150.7]
  Week 36 | -173.8 [-183.5 to -164.1] | -191.5 [-201.1 to -182.0] | -175.6 [-185.2 to -165.9]
  Week 40 | -191.6 [-201.9 to -181.4] | -186.9 [-197.0 to -176.8] | -165.6 [-175.8 to -155.3]
  Week 44 | -181.4 [-191.7 to -171.1] | -188.9 [-199.1 to -178.8] | -177.6 [-187.9 to -167.3]
  Week 48 | -194.5 [-205.1 to -184.0] | -186.8 [-197.1 to -176.6] | -165.8 [-176.3 to -155.4]
  Week 52 | -188.7 [-198.8 to -178.7] | -186.6 [-196.5 to -176.8] | -181.3 [-191.4 to -171.3]
  Week 56 | -196.7 [-207.0 to -186.4] | -189.9 [-200.0 to -179.8] | -174.0 [-184.3 to -163.6]
  Week 60 | -194.3 [-205.6 to -183.0] | -185.2 [-196.3 to -174.1] | -184.1 [-195.5 to -172.7]
  Week 64 | -196.5 [-207.3 to -185.6] | -191.2 [-201.7 to -180.7] | -175.6 [-186.5 to -164.8]
  Week 68 | -194.6 [-204.4 to -184.8] | -192.7 [-202.3 to -183.1] | -186.3 [-196.1 to -176.5]
  Week 72 | -200.9 [-211.0 to -190.8] | -193.4 [-203.3 to -183.5] | -178.0 [-188.1 to -167.9]
  Week 76 | -200.2 [-209.6 to -190.8] | -192.0 [-201.2 to -182.9] | -190.2 [-199.7 to -180.8]
  Week 80 | -202.6 [-212.9 to -192.4] | -190.0 [-199.9 to -180.1] | -182.6 [-192.8 to -172.4]
  Week 84 | -199.3 [-209.8 to -188.7] | -196.0 [-206.3 to -185.8] | -189.5 [-200.0 to -179.0]
  Week 88 | -200.3 [-211.3 to -189.4] | -195.6 [-206.2 to -184.9] | -181.9 [-192.8 to -170.9]
  Week 92 | -199.3 [-209.9 to -188.7] | -196.0 [-206.3 to -185.8] | -187.2 [-197.8 to -176.6]
  Week 96 | -204.5 [-215.1 to -193.8] | -200.8 [-211.1 to -190.4] | -182.9 [-193.5 to -172.2]
  Week 100 | -200.9 [-211.1 to -190.6] | -198.7 [-208.6 to -188.8] | -193.5 [-203.8 to -183.2]

49. Secondary Outcome: Percentage of Participants With Absence of Diabetic Macular Edema in the Study Eye Averaged Over Weeks 48, 52, and 56, ITT and Treatment-Naive Populations
Description: Absence of diabetic macular edema was defined as achieving a central subfield thickness (CST) of <325 microns in the study eye. CST was defined as the distance between the internal limiting membrane and Bruch's membrane. For each participant, an average CST value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Average of Weeks 48, 52, and 56
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 268 | 294 | 279
Percentage of participants
  ITT Population | 85.5 [81.3 to 89.7] | 81.5 [77.1 to 85.9] | 73.2 [68.0 to 78.3]
  Treatment-Naive Population: number analyzed (Participants) | 208 | 232 | 213
  Treatment-Naive Population | 86.0 [81.3 to 90.7] | 83.2 [78.4 to 88.0] | 77.0 [71.3 to 82.6]
Statistical Analysis 1: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 1]; Test type: Other; Difference in CMH Weighted Percentage = 12.3, 95% CI 2-sided [5.7 to 18.9]
Statistical Analysis 2: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 2]; Test type: Other; Difference in CMH Weighted Percentage = 8.2, 95% CI 2-sided [1.5 to 14.9]
Statistical Analysis 3: Comparison: A: Faricimab 6 mg Q8W vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 3]; Test type: Other; Difference in CMH Weighted Percentage = 9.0, 95% CI 2-sided [1.6 to 16.3]
Statistical Analysis 4: Comparison: B: Faricimab 6 mg PTI vs C: Aflibercept 2 mg Q8W; [analysis description as in outcome 23, analysis 4]; Test type: Other; Difference in CMH Weighted Percentage = 6.2, 95% CI 2-sided [-1.2 to 13.6]

50. Secondary Outcome: Percentage of Participants With Absence of Diabetic Macular Edema in the Study Eye Over Time, ITT Population
Description: Absence of diabetic macular edema was defined as achieving a central subfield thickness of <325 microns in the study eye. Central subfield thickness was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 309 | 308 | 308
  Week 4 | 38.2 [32.8 to 43.6] | 43.5 [38.0 to 49.0] | 38.1 [32.8 to 43.5]
  Week 8: number analyzed (Participants) | 304 | 312 | 307
  Week 8 | 53.3 [47.7 to 58.9] | 57.3 [51.9 to 62.7] | 47.9 [42.4 to 53.5]
  Week 12: number analyzed (Participants) | 306 | 304 | 302
  Week 12 | 61.8 [56.5 to 67.2] | 64.8 [59.4 to 70.1] | 56.4 [50.8 to 62.0]
  Week 16: number analyzed (Participants) | 296 | 304 | 294
  Week 16 | 69.2 [64.0 to 74.4] | 69.1 [63.9 to 74.2] | 62.3 [56.8 to 67.8]
  Week 20: number analyzed (Participants) | 294 | 298 | 294
  Week 20 | 73.8 [68.9 to 78.8] | 67.2 [62.0 to 72.4] | 67.4 [62.1 to 72.7]
  Week 24: number analyzed (Participants) | 291 | 302 | 298
  Week 24 | 77.7 [73.0 to 82.4] | 77.9 [73.2 to 82.5] | 62.4 [57.0 to 67.9]
  Week 28: number analyzed (Participants) | 280 | 292 | 286
  Week 28 | 72.1 [67.0 to 77.3] | 81.2 [76.8 to 85.6] | 71.2 [66.1 to 76.4]
  Week 32: number analyzed (Participants) | 277 | 279 | 280
  Week 32 | 80.2 [75.6 to 84.9] | 72.1 [67.0 to 77.3] | 67.0 [61.5 to 72.4]
  Week 36: number analyzed (Participants) | 271 | 279 | 276
  Week 36 | 73.8 [68.7 to 79.0] | 83.8 [79.5 to 88.1] | 74.6 [69.6 to 79.7]
  Week 40: number analyzed (Participants) | 273 | 281 | 275
  Week 40 | 86.1 [82.1 to 90.2] | 81.5 [77.0 to 86.0] | 72.1 [66.9 to 77.3]
  Week 44: number analyzed (Participants) | 269 | 281 | 270
  Week 44 | 81.5 [76.9 to 86.0] | 80.3 [75.7 to 84.9] | 76.6 [71.6 to 81.6]
  Week 48: number analyzed (Participants) | 247 | 281 | 272
  Week 48 | 87.5 [83.4 to 91.6] | 82.7 [78.4 to 87.1] | 71.0 [65.7 to 76.4]
  Week 52: number analyzed (Participants) | 266 | 279 | 271
  Week 52 | 83.7 [79.3 to 88.2] | 82.1 [77.6 to 86.6] | 76.4 [71.5 to 81.4]
  Week 56: number analyzed (Participants) | 263 | 284 | 261
  Week 56 | 89.5 [85.9 to 93.2] | 85.4 [81.4 to 89.5] | 72.2 [66.9 to 77.6]
  Week 60: number analyzed (Participants) | 258 | 273 | 253
  Week 60 | 85.4 [81.1 to 89.6] | 86.1 [82.0 to 90.1] | 78.8 [73.9 to 83.8]
  Week 64: number analyzed (Participants) | 249 | 288 | 258
  Week 64 | 87.6 [83.5 to 91.7] | 82.8 [78.5 to 87.2] | 73.8 [68.5 to 79.0]
  Week 68: number analyzed (Participants) | 252 | 268 | 254
  Week 68 | 85.0 [80.6 to 89.3] | 83.2 [78.8 to 87.6] | 78.2 [73.1 to 83.2]
  Week 72: number analyzed (Participants) | 244 | 260 | 248
  Week 72 | 88.9 [85.1 to 92.8] | 82.4 [77.8 to 86.9] | 74.6 [69.2 to 80.0]
  Week 76: number analyzed (Participants) | 247 | 266 | 247
  Week 76 | 88.4 [84.6 to 92.3] | 82.2 [77.7 to 86.7] | 79.3 [74.3 to 84.4]
  Week 80: number analyzed (Participants) | 243 | 265 | 244
  Week 80 | 90.0 [86.3 to 93.8] | 83.4 [78.9 to 87.8] | 76.6 [71.4 to 81.9]
  Week 84: number analyzed (Participants) | 246 | 261 | 251
  Week 84 | 88.2 [84.2 to 92.2] | 85.8 [81.6 to 90.0] | 80.3 [75.4 to 85.2]
  Week 88: number analyzed (Participants) | 248 | 263 | 245
  Week 88 | 89.5 [85.9 to 93.2] | 85.0 [80.7 to 89.2] | 78.8 [73.8 to 83.9]
  Week 92: number analyzed (Participants) | 246 | 266 | 242
  Week 92 | 88.4 [84.5 to 92.4] | 84.6 [80.3 to 88.9] | 80.3 [75.3 to 85.3]
  Week 96: number analyzed (Participants) | 243 | 263 | 239
  Week 96 | 92.7 [89.5 to 95.8] | 88.1 [84.2 to 92.0] | 80.0 [74.9 to 85.0]
  Week 100: number analyzed (Participants) | 245 | 267 | 233
  Week 100 | 90.6 [87.0 to 94.2] | 85.5 [81.3 to 89.7] | 84.2 [79.6 to 88.8]

51. Secondary Outcome: Percentage of Participants With Retinal Dryness in the Study Eye Over Time, ITT Population
Description: Retinal dryness was defined as achieving a central subfield thickness (ILM-BM) of <280 microns. Central subfield thickness was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. The weighted estimates of the percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world regions were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 4: number analyzed (Participants) | 309 | 308 | 308
  Week 4 | 12.3 [8.7 to 16.0] | 18.5 [14.2 to 22.8] | 15.0 [11.0 to 18.9]
  Week 8: number analyzed (Participants) | 304 | 312 | 307
  Week 8 | 26.2 [21.3 to 31.0] | 25.9 [21.1 to 30.8] | 22.5 [17.9 to 27.2]
  Week 12: number analyzed (Participants) | 306 | 304 | 302
  Week 12 | 33.1 [27.9 to 38.3] | 36.7 [31.3 to 42.0] | 28.2 [23.2 to 33.3]
  Week 16: number analyzed (Participants) | 296 | 304 | 294
  Week 16 | 38.5 [33.1 to 44.0] | 45.0 [39.4 to 50.5] | 33.4 [28.0 to 38.8]
  Week 20: number analyzed (Participants) | 294 | 298 | 294
  Week 20 | 44.3 [38.7 to 49.9] | 41.0 [35.5 to 46.5] | 38.5 [32.9 to 44.0]
  Week 24: number analyzed (Participants) | 291 | 302 | 298
  Week 24 | 50.2 [44.6 to 55.8] | 52.3 [46.8 to 57.9] | 37.0 [31.5 to 42.4]
  Week 28: number analyzed (Participants) | 280 | 292 | 286
  Week 28 | 45.2 [39.5 to 50.8] | 51.9 [46.4 to 57.3] | 46.0 [40.3 to 51.8]
  Week 32: number analyzed (Participants) | 277 | 279 | 280
  Week 32 | 52.3 [46.6 to 58.1] | 46.6 [41.0 to 52.3] | 42.7 [36.9 to 48.4]
  Week 36: number analyzed (Participants) | 271 | 279 | 276
  Week 36 | 50.0 [44.2 to 55.7] | 59.6 [54.0 to 65.1] | 48.8 [42.9 to 54.6]
  Week 40: number analyzed (Participants) | 273 | 281 | 275
  Week 40 | 61.2 [55.5 to 66.8] | 57.7 [52.0 to 63.3] | 49.4 [43.6 to 55.2]
  Week 44: number analyzed (Participants) | 269 | 281 | 270
  Week 44 | 59.9 [54.3 to 65.5] | 58.6 [53.0 to 64.1] | 53.5 [47.7 to 59.4]
  Week 48: number analyzed (Participants) | 247 | 281 | 272
  Week 48 | 67.5 [61.7 to 73.2] | 58.3 [52.8 to 63.8] | 50.2 [44.3 to 56.1]
  Week 52: number analyzed (Participants) | 266 | 279 | 271
  Week 52 | 64.5 [58.8 to 70.1] | 60.9 [55.3 to 66.4] | 54.2 [48.4 to 60.1]
  Week 56: number analyzed (Participants) | 263 | 284 | 261
  Week 56 | 70.3 [64.9 to 75.6] | 63.6 [58.2 to 69.1] | 51.2 [45.2 to 57.1]
  Week 60: number analyzed (Participants) | 258 | 273 | 253
  Week 60 | 65.4 [59.8 to 71.1] | 65.7 [60.1 to 71.2] | 59.2 [53.3 to 65.2]
  Week 64: number analyzed (Participants) | 249 | 288 | 258
  Week 64 | 71.6 [66.2 to 77.1] | 58.7 [53.1 to 64.2] | 52.8 [46.8 to 58.7]
  Week 68: number analyzed (Participants) | 252 | 268 | 254
  Week 68 | 66.9 [61.2 to 72.6] | 60.6 [55.0 to 66.2] | 59.8 [53.9 to 65.8]
  Week 72: number analyzed (Participants) | 244 | 260 | 248
  Week 72 | 71.2 [65.6 to 76.7] | 65.6 [60.1 to 71.1] | 58.8 [52.8 to 64.8]
  Week 76: number analyzed (Participants) | 247 | 266 | 247
  Week 76 | 68.4 [62.9 to 74.0] | 62.8 [57.2 to 68.5] | 58.9 [52.9 to 64.9]
  Week 80: number analyzed (Participants) | 243 | 265 | 244
  Week 80 | 72.6 [67.2 to 78.1] | 64.0 [58.4 to 69.7] | 60.1 [54.1 to 66.1]
  Week 84: number analyzed (Participants) | 246 | 261 | 251
  Week 84 | 68.4 [62.8 to 74.0] | 67.6 [62.1 to 73.1] | 60.7 [54.7 to 66.6]
  Week 88: number analyzed (Participants) | 248 | 263 | 245
  Week 88 | 71.8 [66.4 to 77.2] | 63.3 [57.7 to 68.9] | 60.3 [54.2 to 66.4]
  Week 92: number analyzed (Participants) | 246 | 266 | 242
  Week 92 | 72.9 [67.5 to 78.3] | 64.6 [59.0 to 70.2] | 64.0 [58.0 to 70.1]
  Week 96: number analyzed (Participants) | 243 | 263 | 239
  Week 96 | 75.1 [69.9 to 80.3] | 67.4 [62.0 to 72.9] | 63.1 [57.0 to 69.1]
  Week 100: number analyzed (Participants) | 245 | 267 | 233
  Week 100 | 72.0 [66.6 to 77.4] | 69.3 [63.9 to 74.6] | 64.8 [58.8 to 70.9]

52. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye Over Time, ITT Population
Description: Intraretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world); Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 48, 52, 56, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 16: number analyzed (Participants) | 296 | 303 | 294
  Week 16 | 19.6 [15.1 to 24.1] | 19.8 [15.4 to 24.2] | 13.3 [9.4 to 17.1]
  Week 48: number analyzed (Participants) | 246 | 276 | 269
  Week 48 | 40.9 [34.8 to 47.0] | 32.3 [26.9 to 37.7] | 22.5 [17.6 to 27.3]
  Week 52: number analyzed (Participants) | 262 | 280 | 269
  Week 52 | 39.1 [33.3 to 44.9] | 35.9 [30.3 to 41.5] | 28.4 [23.1 to 33.7]
  Week 56: number analyzed (Participants) | 260 | 277 | 258
  Week 56 | 42.5 [36.6 to 48.3] | 39.9 [34.2 to 45.6] | 27.3 [22.0 to 32.7]
  Week 92: number analyzed (Participants) | 240 | 259 | 234
  Week 92 | 56.0 [49.8 to 62.2] | 45.0 [39.0 to 51.0] | 39.2 [33.0 to 45.4]
  Week 96: number analyzed (Participants) | 239 | 256 | 231
  Week 96 | 62.3 [56.3 to 68.4] | 47.6 [41.5 to 53.6] | 39.1 [32.8 to 45.3]
  Week 100: number analyzed (Participants) | 238 | 261 | 229
  Week 100 | 56.6 [50.4 to 62.8] | 52.2 [46.2 to 58.1] | 45.1 [38.7 to 51.4]

53. Secondary Outcome: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye Over Time, ITT Population
Description: Subretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world); Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 48, 52, 56, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 16: number analyzed (Participants) | 294 | 305 | 293
  Week 16 | 99.0 [97.9 to 100.0] | 96.7 [94.7 to 98.7] | 95.6 [93.3 to 97.8]
  Week 48: number analyzed (Participants) | 251 | 280 | 272
  Week 48 | 97.2 [95.1 to 99.2] | 95.8 [93.5 to 98.1] | 95.3 [92.8 to 97.8]
  Week 52: number analyzed (Participants) | 267 | 281 | 271
  Week 52 | 94.7 [91.9 to 97.4] | 95.7 [93.4 to 98.0] | 97.8 [96.1 to 99.5]
  Week 56: number analyzed (Participants) | 266 | 283 | 263
  Week 56 | 97.0 [95.0 to 99.0] | 95.8 [93.5 to 98.1] | 95.9 [93.5 to 98.2]
  Week 92: number analyzed (Participants) | 245 | 264 | 241
  Week 92 | 95.0 [92.3 to 97.8] | 96.2 [93.9 to 98.5] | 96.0 [93.5 to 98.4]
  Week 96: number analyzed (Participants) | 244 | 263 | 238
  Week 96 | 96.3 [94.0 to 98.7] | 96.6 [94.5 to 98.8] | 96.2 [93.8 to 98.6]
  Week 100: number analyzed (Participants) | 247 | 266 | 233
  Week 100 | 96.0 [93.5 to 98.4] | 96.2 [93.9 to 98.5] | 95.9 [93.5 to 98.3]

54. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye Over Time, ITT Population
Description: Intraretinal fluid and subretinal fluid were measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥64 vs. <64 letters), prior IVT anti-VEGF therapy (yes vs. no), and region (U.S. and Canada vs. rest of the world); Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 16, 48, 52, 56, 92, 96, and 100
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
Percentage of participants
  Week 16: number analyzed (Participants) | 296 | 303 | 294
  Week 16 | 19.6 [15.1 to 24.1] | 19.1 [14.8 to 23.5] | 13.3 [9.4 to 17.1]
  Week 48: number analyzed (Participants) | 246 | 276 | 269
  Week 48 | 40.5 [34.4 to 46.6] | 31.2 [25.8 to 36.6] | 22.5 [17.6 to 27.3]
  Week 52: number analyzed (Participants) | 262 | 279 | 269
  Week 52 | 39.1 [33.3 to 44.9] | 34.9 [29.4 to 40.5] | 28.4 [23.1 to 33.7]
  Week 56: number analyzed (Participants) | 261 | 277 | 258
  Week 56 | 42.3 [36.4 to 48.2] | 39.2 [33.5 to 44.9] | 26.6 [21.3 to 31.8]
  Week 92: number analyzed (Participants) | 240 | 259 | 234
  Week 92 | 55.2 [49.0 to 61.4] | 44.2 [38.2 to 50.2] | 38.3 [32.2 to 44.5]
  Week 96: number analyzed (Participants) | 239 | 256 | 231
  Week 96 | 61.0 [54.9 to 67.2] | 46.5 [40.4 to 52.5] | 38.2 [32.0 to 44.4]
  Week 100: number analyzed (Participants) | 238 | 262 | 228
  Week 100 | 54.9 [48.7 to 61.2] | 51.2 [45.2 to 57.2] | 44.8 [38.4 to 51.2]

55. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) Composite Score Over Time, ITT Population
Description: The NEI VFQ-25 captures a patient's perception of vision-related functioning and quality of life. The core measure includes 25 items that comprise 11 vision-related subscales and one item on general health. The composite score ranges from 0 to 100, with higher scores, or a positive change from baseline, indicating better vision-related functioning. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline NEI VFQ-25 Composite Score (continuous), baseline BCVA (<64 vs. ≥64 letters), prior intravitreal anti-VEGF therapy (yes vs. no), and region of enrollment. An unstructured covariance structure was used. Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% CI is a rounding of 95.04% CI.
Time Frame: Baseline, Weeks 24, 52, and 100
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 315
score on a scale
  Week 24 | 5.7 [4.6 to 6.9] | 6.5 [5.4 to 7.7] | 7.0 [5.9 to 8.1]
  Week 52 | 6.8 [5.5 to 8.2] | 6.6 [5.3 to 7.9] | 7.6 [6.3 to 9.0]
  Week 100 | 8.8 [7.3 to 10.3] | 7.3 [5.9 to 8.7] | 6.9 [5.4 to 8.4]

56. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: This analysis of adverse events (AEs) includes both ocular and non-ocular (systemic) AEs. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. AEs of special interest included the following: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law; Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation.
Time Frame: From first dose of study drug through end of study (up to 2 years)
Population: The safety-evaluable population comprised all participants who received at least one injection of active study drug (faricimab or aflibercept) in the study eye.
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 314
Percentage of participants
  Adverse Event (AE) | 89.3 | 85.3 | 87.3
  Serious AE (SAE) | 30.6 | 25.7 | 31.8
  AE Leading to Withdrawal from Study Treatment | 2.2 | 2.8 | 1.6
  AE of Special Interest (AESI) | 7.6 | 7.2 | 6.4

57. Secondary Outcome: Percentage of Participants With at Least One Ocular Adverse Event in the Study Eye or the Fellow Eye
Description: This analysis of adverse events (AEs) only includes ocular AEs, which are categorized as having occurred either in the study eye or the fellow eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: From first dose of study drug through end of study (up to 2 years)
Population: as for outcome 56
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 314
Percentage of participants
  Study Eye: Adverse Event (AE) | 52.4 | 51.7 | 44.6
  Study Eye: Serious AE (SAE) | 4.4 | 6.3 | 4.1
  Study Eye: AE Leading to Withdrawal from Treatment | 0.3 | 1.9 | 0.3
  Study Eye: Treatment-related AE | 3.2 | 4.4 | 4.8
  Study Eye: Treatment-related SAE | 0.0 | 0.9 | 0.0
  Study Eye: AE of Special Interest (AESI) | 4.4 | 6.3 | 3.8
  Study Eye: AESI, Drop in Visual Acuity (VA) Score ≥30 Letters | 3.2 | 5.0 | 2.9
  Study Eye: AESI, Associated with Severe Intraocular Inflammation (IOI) | 0.3 | 0.0 | 0.3
  Study Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 0.9 | 1.3 | 1.0
  Fellow Eye: AE | 50.5 | 43.3 | 44.3
  Fellow Eye: SAE | 3.5 | 1.9 | 3.5
  Fellow Eye: AESI | 3.8 | 0.9 | 2.9
  Fellow Eye: AESI, Drop in VA Score ≥30 Letters | 3.5 | 0.6 | 2.5
  Fellow Eye: AESI, Associated with Severe IOI | 0.0 | 0.0 | 0.0
  Fellow Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 0.3 | 0.3 | 0.3

58. Secondary Outcome: Percentage of Participants With at Least One Non-Ocular Adverse Event
Description: This analysis of adverse events (AEs) only includes non-ocular (systemic) AEs. Investigators sought information on adverse events (AEs) at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. The non-ocular AE of special interest was: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From first dose of study drug through end of study (up to 2 years)
Population: as for outcome 56
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
Number analyzed (Participants) | 317 | 319 | 314
Percentage of participants
  Adverse Event (AE) | 69.4 | 68.3 | 73.6
  Serious AE (SAE) | 24.0 | 20.1 | 28.3
  AE Leading to Withdrawal from Study Treatment | 1.9 | 0.9 | 1.3
  AE of Special Interest (AESI) | 0.0 | 0.0 | 0.0

59. Secondary Outcome: Plasma Concentration of Faricimab Over Time
Description: Faricimab concentration in plasma was determined using a validated immunoassay method.
Time Frame: Pre-dose on Day 1 (Baseline); Weeks 4, 28, 52, 76, and 100
Population: This analysis only included participants in Arms A and B who received treatment with faricimab and with at least one plasma sample, provided sufficient dosing information (dose and dosing time) was available. The number of participants analyzed at a given timepoint includes those with an available plasma sample and dosing information at that timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 315 | 319
micrograms per millilitre (μg/mL)
  Baseline: number analyzed (Participants) | 298 | 305
  Baseline | 0.0001 (0.0020) | 0.0000 (0.0004)
  Week 4: number analyzed (Participants) | 284 | 287
  Week 4 | 0.0192 (0.0163) | 0.0196 (0.0151)
  Week 28: number analyzed (Participants) | 266 | 283
  Week 28 | 0.0030 (0.0050) | 0.0115 (0.0189)
  Week 52: number analyzed (Participants) | 248 | 270
  Week 52 | 0.0042 (0.0078) | 0.0113 (0.0140)
  Week 76: number analyzed (Participants) | 237 | 250
  Week 76 | 0.0060 (0.0093) | 0.0060 (0.0103)
  Week 100: number analyzed (Participants) | 254 | 267
  Week 100 | 0.0058 (0.0106) | 0.0071 (0.0110)

60. Secondary Outcome: Percentage of Participants Who Test Positive for Treatment-Emergent Anti-Drug Antibodies Against Faricimab During the Study
Description: Anti-drug antibodies (ADAs) against fariciamb were detected in plasma using a validated bridging enzyme-linked immunosorbent assay (ELISA). The percentage of participants with treatment-emergent ADA-positive samples includes post-baseline evaluable participants with at least one treatment-induced (defined as having an ADA-negative sample or missing sample at baseline and any positive post-baseline sample) or treatment-boosted (defined as having an ADA-positive sample at baseline and any positive post-baseline sample with a titer that is equal to or greater than 4-fold baseline titer) ADA-positive sample during the study treatment period.
Time Frame: Baseline, Weeks 4, 28, 52, 76, and 100
Population: The analysis population consisted of all participants receiving faricimab with at least one determinant post-baseline ADA assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI
Number analyzed (Participants) | 313 | 318
Percentage of participants
  Total Treatment-Emergent ADA-Positive | 7.0 | 8.2
  Treatment-Induced ADA-Positive | 7.0 | 8.2
  Treatment-Boosted ADA-Positive | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From Baseline until Week 100
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For ocular AEs, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Arm/Group | A: Faricimab 6 mg Q8W | B: Faricimab 6 mg PTI | C: Aflibercept 2 mg Q8W
All-Cause Mortality (participants affected / at risk) | 12/317 | 9/319 | 10/314
Serious Adverse Events (participants affected / at risk) | 97/317 | 82/319 | 100/314
Other Adverse Events (participants affected / at risk) | 195/317 | 169/319 | 178/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Faricimab 6 mg Q8W (N=317) | B: Faricimab 6 mg PTI (N=319) | C: Aflibercept 2 mg Q8W (N=314)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 3 (3)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (5) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 3 (4) | 4 (5)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 8 (10) | 4 (5) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Subendocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 4 (5) | 7 (7) | 7 (7)
Cataract subcapsular (Eye disorders) | 1 (2) | 1 (1) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 7 (10) | 2 (2) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 2 (2) | 3 (4)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 1 (2)
Retinal tear (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 4 (4) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 3 (4) | 1 (1) | 8 (8)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gallbladder empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (2) | 2 (4) | 1 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (2) | 3 (4)
Pneumonia (Infections and infestations) | 7 (7) | 6 (6) | 5 (6)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (6)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic endorgan damage (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (7)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 4 (4) | 4 (5)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 0 (0) | 3 (3)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperplasia adrenal (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic eye disease (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal varices (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 7 (8) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Biopsy bladder (Investigations) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemodialysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Faricimab 6 mg Q8W (N=317) | B: Faricimab 6 mg PTI (N=319) | C: Aflibercept 2 mg Q8W (N=314)
Cataract (Eye disorders) | 52 (77) | 58 (88) | 33 (48)
Conjunctival haemorrhage (Eye disorders) | 36 (44) | 24 (29) | 25 (34)
Diabetic retinal oedema (Eye disorders) | 29 (31) | 25 (30) | 23 (27)
Vitreous detachment (Eye disorders) | 19 (26) | 18 (21) | 27 (30)
Nasopharyngitis (Infections and infestations) | 30 (35) | 27 (34) | 38 (43)
Urinary tract infection (Infections and infestations) | 14 (20) | 15 (18) | 27 (35)
Headache (Nervous system disorders) | 18 (36) | 11 (16) | 8 (10)
Hypertension (Vascular disorders) | 20 (22) | 26 (29) | 16 (16)
Dry eye (Eye disorders) | 19 (34) | 22 (39) | 11 (24)
Vitreous floaters (Eye disorders) | 17 (22) | 12 (15) | 18 (21)
Fall (Injury, poisoning and procedural complications) | 18 (23) | 8 (8) | 14 (19)
Intraocular pressure increased (Investigations) | 21 (34) | 14 (23) | 15 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 7 (7) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 16 (17) | 10 (10)

LIMITATIONS AND CAVEATS:
All secondary outcome measures were unpowered for statistical analysis, and the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03622593/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT03622593/SAP_001.pdf